#### The GlaxoSmithKline group of companies

| Division | : | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | : | Reporting and Analysis Plan (RAP) |

Title : Reporting and Analysis Plan for an open-label study to evaluate correct use and ease of use of the ELLIPTA Dry Powder Inhaler (DPI) in pediatric patients currently receiving inhaled therapy for treatment of their asthma

Compound Number : GSK2285997 (GW685698 + GW642444)

Effective Date : 12-MAR-2019

#### **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 206924.
- This RAP is intended to describe the planned analyses required for the study and output to be included in the Clinical Study Report for Protocol 206924.
- This RAP will be provided to the study team members to convey the content of the Statistical Analysis Complete (SAC) deliverable.

#### **RAP Author(s):**

| Author | | Date |
|--------------|-----------------------------------|-------------|
| Lead | | |
| PPD | | 06-MAR-2019 |
| Statistician | (Respiratory Clinical Statistics) | |

Copyright 2019 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

# **RAP Team Review Confirmations (Method: E-mail):**

| Reviewer(s | Date | |
|-------------|---------------------------------------|--------------|
| PPD | (review confirmation on behalf of PPD | |
| Clinical De | 07-MAR-2019 | |
| Developmen | nt) | |
| PPD | | 07 MAD 2010 |
| Programmin | 07-MAR-2019 | |
| PPD | | 08-MAR-2019 |
| Associate N | Ianager (Biostatistics) | U0-WIAK-2019 |

# Clinical Statistics and Clinical Programming Line Approvals (Method: Pharma TMF eSignature):

| Approver(s) | Date |
|--------------------------------------------------------------|-------------|
| Senior Statistics Director (Respiratory Clinical Statistics) | 08-MAR-2019 |
| Programming Manager (Respiratory Clinical Programming) | 12-MAR-2019 |

# **TABLE OF CONTENTS**

| | | | | | PAGE |
|---|---|---|---|---|---|
| 1. | INTRO | DDUCTIO | N | | 8 |
| 2. | CLIMAN | MDV OF | KEN DDU. | TOCOL INFORMATION | Ω |
| ۷. | 2.1. | | | otocol Defined Statistical Analysis Plan | |
| | 2.1. | | | | |
| | 2.2. | | | and Endpoint(s) | |
| | 2.3.<br>2.4. | | | ses / Statistical Analyses | |
| | 2.4. | Statistica | аг пуроше | ses / Statistical Arialyses | |
| 3. | PLAN | NED ANA | LYSES | | 12 |
| | 3.1. | Interim A | Analyses | | 12 |
| | 3.2. | Final An | alyses | | 12 |
| 4 | ANAI | YSIS POF | PUI ATION | S | 12 |
| •• | 4.1. | | | S | |
| | т. г. | 1 1010001 | Deviations | <b>,</b> | |
| 5. | | | | DATA ANALYSES AND DATA HANDLING | 4.4 |
| | | | | O.b. married District Descriptions | |
| | 5.1. | | | Sub-group Display Descriptors | |
| | 5.2. | | | S | |
| | 5.3. | | | ) | |
| | 5.4. | | | variates, Other Strata and Subgroups | |
| | | 5.4.1. | | es and Other Strata | |
| | | 5.4.2. | | ion of Subgroups | |
| | 5.5. | | | ons and Multiplicity | 15 |
| | 5.6. | | | ns for Data Analyses and Data Handling | 15 |
| 6. | | | | IALYSES | |
| | 6.1. | | | ed Study Population Analyses | |
| | 6.2. | | | tion | |
| | 6.3. | Medical | Conditions | | 16 |
| | 6.4. | Concom | itant Medic | cations | 16 |
| | 6.5. | Incorrect | t Use at Vi | sit 1 | 17 |
| 7. | FFFIC | CACY AND | N YSES | | 18 |
| | 7.1. | | | nalyses | |
| | 7.1. | 7.1.1. | • | S | |
| | | 7.1.1.<br>7.1.2. | | Measure | |
| | | 7.1.2.<br>7.1.3. | | n of Interest | |
| | | 7.1.3.<br>7.1.4. | | for Intercurrent (Post-Randomization) Events | |
| | | 7.1. <del>4</del> . | 7.1.4.1. | , | 10 |
| | | | 7.1.4.1. | Percentage of participants from each stratum who demonstrate correct use of the ELLIPTA | |
| | | | | | 10 |
| | | | 7110 | DPI after the study period at V2 | 19 |
| | | | 7.1.4.2. | Percentage of participants from each stratum | |
| | | | | who rate the ELLIPTA DPI as easy to use, | |
| | | | | from those who could demonstrate correct use | |
| | | | | of the ELLIPTA DPI after the study period at | 4.0 |
| | | | | V2 | 19 |


| 206924 |
|--------|

| | 7.1.5. | Statistical | Analyses / N | /lethods | 20 |
|---|---|---|---|---|---|
| | | 7.1.5.1. | Statistical N | Methodology Specification | 20 |
| | | | 7.1.5.1.1. | | |
| | | | | each stratum who demonstrate | |
| | | | | correct use of the ELLIPTA DPI | |
| | | | | after the study period at V2 | 20 |
| | | | 7.1.5.1.2. | • • | |
| | | | | each stratum who rate the | |
| | | | | ELLIPTA DPI as easy to use, from | |
| | | | | those who could demonstrate | |
| | | | | correct use of the ELLIPTA DPI | |
| | | | | after the study period at V2 | 21 |
| 7.2. | Seconda | | | | |
| | 7.2.1. | | | | |
| | 7.2.2. | Summary | Measure | | 22 |
| | 7.2.3. | Populatio | n of Interest. | | 22 |
| | 7.2.4. | Strategy f | or Intercurre | nt (Post-Randomization) Events | 22 |
| | | 7.2.4.1. | Percentage | e of participants from each stratum | |
| | | | | nstrate correct use of the ELLIPTA | |
| | | | | itial training from HCP at V1 | 22 |
| | | 7.2.4.2. | | e of participants who demonstrate | |
| | | | | of the ELLIPTA DPI after the study | |
| | | | | 2 | 23 |
| | | 7.2.4.3. | | e of participants who rate the | |
| | | 7.2.1.0. | | PI as easy to use, from those who | |
| | | | | onstrate correct use of the ELLIPTA | |
| | | | | e study period at V2 | 23 |
| | | 7.2.4.4. | | e of participants from each stratum | 20 |
| | | 7.2.4.4. | | at least one critical error during use | |
| | | | | PTA DPI after initial training from | |
| | | | | | 24 |
| | 7.2.5. | Statistical | | | |
| | 7.2.5. | | | Methods | |
| | | 7.2.5.1. | | Methodology Specification | 25 |
| | | | 7.2.5.1.1. | 9 1 1 | |
| | | | | each stratum who demonstrate | |
| | | | | correct use of the ELLIPTA DPI | |
| | | | | after initial training from HCP at | |
| | | | | V1 | 25 |
| | | | 7.2.5.1.2. | Percentage of participants who | |
| | | | | demonstrate correct use of the | |
| | | | | ELLIPTA DPI after the study | |
| | | | | period at V2 | 25 |
| | | | 7.2.5.1.3. | Percentage of participants who | |
| | | | | rate the use of the ELLIPTA DPI | |
| | | | | as easy to use, from those who | |
| | | | | could demonstrate correct use of | |
| | | | | the ELLIPTA DPI after the study | |
| | | | | period at V2 | 26 |
| | | | 7.2.5.1.4. | Percentage of participants from | |
| | | | | each stratum who made at least | |
| | | | | one critical error during use of the | |
| | | | | <b>5</b> | |

| | | | | ELLIPTA DPI after initial training | 00 |
|---|---|---|---|---|---|
| 7.3. | Evolora | ton, Efficac | v Analyses | from HCP at V1 | |
| 1.5. | 7.3.1. | • | • | | |
| | 7.3.2. | | | | |
| | 7.3.3. | | | | |
| | 7.3.4. | | | nt (Post-Randomization) Events | |
| | | 7.3.4.1. | | e of participants from each stratum | 20 |
| | | | ne ability to tell how many puffs are | | |
| | | | ELLIPTÁ DPI as easy after the study | | |
| | | | | ′2 | 28 |
| | | 7.3.4.2. | Percentage | e of participant's parents/guardians | |
| | | | who rate th | ne ability to tell how many doses are | |
| | | | | in the ELLIPTA DPI as easy or very | |
| | | | | the study period at V2 | 29 |
| | | 7.3.4.3. | | e of participant's parents/guardians | |
| | | | | be likely or very likely to ask their | |
| | | | | he ELLIPTA DPI if the participants | |
| | | | | ly inhaled medication(s) were | |
| | | | the ELLIPTA DPI after the study | 00 | |
| | | 7.3.4.4. | | 2e of participants from each stratum | 30 |
| | | 7.3.4.4. | _ | nstrate correct use after the study | |
| | | | 2 with assistance from | | |
| | | | ardians | 30 | |
| | | 7.3.4.5. | | e of participants from each stratum | |
| | | | | at least one critical error during use | |
| | | | | PTA DPI after the study period at | |
| | | | | | 31 |
| | | 7.3.4.6. | Percentage | e of participants who made at least | |
| | | | | error during use of the ELLIPTA | |
| | | | | nitial training from HCP at V1 | |
| | 7.3.5. | | | Methods | |
| | | 7.3.5.1. | | Methodology Specification | 32 |
| | | | 7.3.5.1.1. | Percentage of participants from | |
| | | | | each stratum who rate the ability | |
| | | | | to tell how many puffs are left in | |
| | | | | the ELLIPTA DPI as easy after the study period at V2 | 20 |
| | | | 7.3.5.1.2. | study period at V2 Percentage of participant's | 32 |
| | | | 1.3.3.1.2. | parents/guardians who rate the | |
| | | | | ability to tell how many doses are | |
| | | | | remaining in the ELLIPTA DPI as | |
| | | | | easy or very easy after the study | |
| | | | | period at V2 | 33 |
| | | | 7.3.5.1.3. | Percentage of participant's | |
| | | | | parents/guardians who would be | |
| | | | | likely or very likely to ask their | |
| | | | | doctor for the ELLIPTA DPI if the | |
| | | | | participants current daily inhaled | |
| | | | | medication(s) were available in | |

| | | | | the ELLIPTA DPI after the study | |
|---|---|---|---|---|---|
| | | | | period at V2 | 33 |
| | | | 7.3.5.1.4. | Percentage of participants from | |
| | | | | each stratum who demonstrate | |
| | | | | correct use after the study period | |
| | | | | at V2 with assistance from | 0.4 |
| | | | 70545 | parents/guardians | 34 |
| | | | 7.3.5.1.5. | Percentage of participants from | |
| | | | | each stratum who made at least | |
| | | | | one critical error during use of the | |
| | | | | ELLIPTA DPI after the study | 25 |
| | | | 72516 | period at V2. | 35 |
| | | | 7.3.5.1.6. | Percentage of participants who | |
| | | | | made at least one critical error | |
| | | | | during use of the ELLIPTA DPI | |
| | | | | after initial training from HCP at V1 | 25 |
| | | | | V 1 | 30 |
| 8. | SAFET | γ ΔΝΔΙ γ | SES | | 36 |
| 0. | 8.1. | | | | |
| | 8.2. | | | est Analyses | |
| | 0.2. | / laverse | Events of openial intere | 55t / Wary 505 | |
| 9. | REFE | RENCES | | | 37 |
| 10. | APPE | NDICES | | | 38 |
| | 10.1. | Appendix | 1: Protocol Deviation N | Management | 38 |
| | | | | rotocol Population | |
| | 10.2. | | | es | |
| | | 10.2.1. | Protocol Defined Sche | dule of Events | 39 |
| | 10.3. | | | ws | |
| | | | | ent Windows for Analyses | 41 |
| | 10.4. | | | Freatment Emergent Adverse | |
| | | 10.4.1. | | | |
| | | | | es for Concomitant Medication | |
| | | 10.4.2. | | lag for Adverse Events | |
| | 10.5. | | | ards & Handling Conventions | |
| | | 10.5.1. | | | |
| | 40.0 | 10.5.2. | | | |
| | 10.6. | | | ormed Data | |
| | | 10.6.1. | | | |
| | | 10.6.2. | | | |
| | | 10.6.3.<br>10.6.4. | | | |
| | 10.7 | | | o for Missian Data | |
| | 10.7. | | | s for Missing Data | |
| | | 10.7.1. | | S | |
| | | 10.7.2. | | ata Missing and Partial Dates | |
| | 10.8. | Annendiv | | Clinical Importance | |
| | 10.0. | 10.8.1. | | Cililical Importance | |
| | 10.9. | | | de Marks | |
| | 10.5. | | | ue iviai ks | |
| | | | , was a ridual to | | |


| 10.9.2. Trademarks | 51 |
|-----------------------------------------------------------|------------------|
| 10.10. Appendix 10: List of Data Displays | 5 <mark>2</mark> |
| 10.10.1. Data Display Numbering | |
| 10.10.2. Mock Example Shell Referencing | 52 |
| 10.10.3. Deliverables | 52 |
| 10.10.4. Study Population Tables | 53 |
| 10.10.5. Efficacy Tables | 57 |
| 10.10.6. Efficacy Figures | 60 |
| 10.10.7. Safety Tables | 62 |
| 10.10.8. ICH Listings | 64 |
| 10.10.9. Non-ICH Listings | 68 |
| 10.11. Appendix 11: Example Mock Shells for Data Displays | |

### 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Study Report for Protocol: 206924.

| Revision Chronology | : | |
|---------------------|-------------|----------|
| 2017N346371_00 | 23-JAN-2018 | Original |

#### 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

Changes from the originally planned statistical analysis specified in the protocol (dated: 23/JAN/2018) are outlined in Table 1.

Table 1 Changes to Protocol Defined Analysis Plan

| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Statistical Analysis Plan | Statistical Analysis Plan | Rationale for Changes |
| Protocol Section 10.3 Populations for Analyses | RAP Section 4 Analysis<br>Populations | The analysis populations have been updated to follow the study populations standard definitions and statistical displays |
| | RAP Section 7.1.5.1.2, Section 7.2.5.1.3., Section 7.3.4.1. | Removed sensitivity analysis proposed in the critical components RAP "participants who completed demonstration of correct use before answering the ease of use questionnaire" due to the information not being recorded. |

# 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| To determine the proportion of participants<br>from each stratum who demonstrate correct<br>use of the ELLIPTA DPI after the study period<br>at V2. | The percentage of participants from each<br>stratum who demonstrate correct use of the<br>ELLIPTA DPI after the study period at V2. |
| To determine the proportion of participants from each stratum who rate the use of the ELLIPTA DPI as easy to use, from those who could demonstrate correct use of the ELLIPTA DPI after the study period at V2. | The percentage of participants from each stratum who rate the ELLIPTA DPI as easy to use, from those who could demonstrate correct use of the ELLIPTA DPI after the study period at V2. |

| Objectives Endpoints | | |
|---|---|---|
| Secondary Objectives | | Secondary Endpoints |
| To determine the proportion<br>from each stratum who der<br>use of the ELLIPTA DPI aft<br>from healthcare profession. | n of participants<br>monstrate correct<br>ter initial training | The percentage of participants from each<br>stratum who demonstrate correct use of the<br>ELLIPTA DPI after initial training from HCP at<br>V1. |
| To determine the proportion<br>demonstrate correct use of<br>after the study period at V2 | n of participants who the ELLIPTA DPI | <ul> <li>The percentage of participants who demonstrate<br/>correct use of the ELLIPTA DPI after the study<br/>period at V2.</li> </ul> |
| To determine the proportion rate the use of the ELLIPTA use, from those who could use of the ELLIPTA DPI aft at V2. | A DPI as easy to demonstrate correct | <ul> <li>The percentage of participants who rate the<br/>ELLIPTA DPI as easy to use, from those who<br/>could demonstrate correct use of the ELLIPTA<br/>DPI after the study period at V2.</li> </ul> |
| To determine the proportion<br>from each stratum who may<br>critical error during use of the<br>after initial training from HC | de at least one<br>he ELLIPTA DPI<br>CP at V1. | <ul> <li>The percentage of participants from each<br/>stratum who made at least one critical error<br/>during use of the ELLIPTA DPI after initial<br/>training from HCP at V1.</li> </ul> |
| Exploratory Objectives | | Exploratory Endpoints |
| <ul> <li>To determine the proportion from each stratum who rate how many puffs are left in the easy after the study period</li> <li>To determine the proportion parents/guardians who rate</li> </ul> | e the ability to tell the ELLIPTA DPI as at V2. n of participant's | <ul> <li>The percentage of participants from each stratum who rate the ability to tell how many puffs are left in the ELLIPTA DPI as easy after the study period at V2.</li> <li>The percentage of participant's parents/guardians who rate the ability to tell how</li> </ul> |
| how many doses are remain DPI as 'easy 'or 'very easy' period at V2. | ining in the ELLIPTA | many doses are remaining in the ELLIPTA DPI as 'easy' or 'very easy' after the study period at V2. |
| To determine the proportion parents/guardians who wou 'very likely' to ask their doc DPI if the participants curre medication(s) were availab DPI after the study period as | uld be 'likely' or<br>tor for the ELLIPTA<br>ent daily inhaled<br>le in the ELLIPTA | <ul> <li>The percentage of participant's<br/>parents/guardians who would be 'likely' or<br/>'very likely' to ask their doctor for the ELLIPTA<br/>DPI if the participants current daily inhaled<br/>medication(s) were available in the ELLIPTA DPI<br/>after the study period at V2.</li> </ul> |
| To determine the proportion<br>from each stratum who can<br>correct use after the study<br>assistance from parents/gu | n demonstrate<br>period at V2 with | <ul> <li>The percentage of participants from each<br/>stratum who demonstrated correct use after the<br/>study period at V2 with assistance from<br/>parents/guardians.</li> </ul> |
| To determine the proportion<br>from each stratum who man<br>critical error during use of the<br>after the study period at V2 | de at least one<br>he ELLIPTA DPI | <ul> <li>The percentage of participants from each<br/>stratum who made at least one critical error<br/>during use of the ELLIPTA DPI after the study<br/>period at V2.</li> </ul> |
| To determine the proportion<br>made at least one critical e<br>the ELLIPTA DPI after initia<br>at V1. | rror during use of | <ul> <li>The percentage of participants who made at<br/>least one critical error during use of the ELLIPTA<br/>DPI after initial training from HCP at V1.</li> </ul> |

## 2.3. Study Design



# 2.4. Statistical Hypotheses / Statistical Analyses

This is a descriptive, placebo only study and no formal inference is planned. The two primary objectives of the study are:

- To determine the proportion of participants from each stratum who demonstrate correct use of the ELLIPTA DPI after the study period at V2.
- To determine the proportion of participants from each stratum who rate the use of the ELLIPTA DPI as easy to use, from those who could demonstrate correct use of the ELLIPTA DPI after the study period at V2.

### 3. PLANNED ANALYSES

## 3.1. Interim Analyses

No interim analysis is planned for this study.

# 3.2. Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- 1. All participants have completed the study as defined in the protocol.
- 2. All required database cleaning activities have been completed and final database release (DBR) and database freeze (DBF) has been declared by Data Management.
- 3. All criteria for unblinding the randomization codes have been met.
- 4. Randomization codes have been distributed according to RandAll NG procedures.

#### 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| All Subjects<br>Enrolled (ASE) | All participants whose parent/guardian has signed the Informed Consent Form (ICF) and the accompanying informed assent from the participant (where applicable) has been acquired, and for whom a record exists in the study database, including screen failures and any participant who was not screened but experienced an SAE between the date of informed consent and the planned date of the Screening visit. | <ul><li>Study Population</li><li>Safety</li></ul> |
| Intent-To-Treat<br>(ITT) | The Intent-to-Treat (ITT) population is defined as all subjects who have been screened and received at least one dose of the study medication (placebo). | <ul><li>Study Population</li><li>Safety</li><li>Efficacy</li></ul> |
| Modified Intent-<br>to-Treat<br>(MITT) | The Modified Intent-to-Treat (MITT) population is defined as all subjects who have been screened, received at least one dose of the study medication (placebo) and were randomized to a version of the ease of use questionnaire at V2. | Study Population Efficacy |

Refer to Appendix 10: List of Data Displays which details the population used for each display. – Appendix 10 to be defined in full RAP

#### 4.1. Protocol Deviations

Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.


206924

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan 8-JUN-2018, Version 1.0.

- o Data will be reviewed prior to freezing the database to ensure all important deviations are captured and categorised on the protocol deviations dataset.
- This dataset will be the basis for the summaries and listings of protocol deviations.

A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the eCRF.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

## 5.1. Study Treatment & Sub-group Display Descriptors

All participants during screening will be provided an ELLIPTA DPI placebo to demonstrate correct use at Visit 1 at site and provided another ELLIPTA DPI to take away from site for the study period. The ELLIPTA DPI placebo is the only 'treatment' being provided in this study, hence no formal treatment comparisons will be performed.

All participants will be stratified in to two strata based on their age at visit 0 (5-7 and 8-11 years old).

The participants who make it through visit 1 and return at visit 2 will be randomised to one of two ELLIPTA DPI ease of use questionnaires (version A or version B). The version of the ease of use questionnaires will be considered the "treatment groups" in this study. The parents/guardians are also assigned to one of two ease of use questionnaires. The participant's questions are different to the parents/guardian's versions, however, the parents/guardians are assigned the same version (A or B) as their child's randomised version.

| | Treatment Group Descriptions | | |
|---|---|---|---|
| RandAll NG Data Displays for Reporting | | Reporting | |
| Code | Description | Description | Order in TLF |
| A | Placebo Ease of Use Questionnaire Version A | Questionnaire: Version A | 1 |
| В | Placebo Ease of Use Questionnaire Version B | Questionnaire: Version B | 2 |

### 5.2. Baseline Definitions

For all endpoints, the baseline value will be the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. If time is not collected, Day 1 assessments are assumed to be taken prior to first dose and used as baseline.

Unless otherwise stated, if baseline data is missing no derivation will be performed and baseline will be set to missing.

#### 5.3. Multicentre Studies

In this multicentre global study, enrolment will be presented by country.

| Region | Countries |
|------------------|-----------------------|
| Northern America | United States, Canada |

## 5.4. Examination of Covariates, Other Strata and Subgroups

#### 5.4.1. Covariates and Other Strata

The list of covariates and other strata may be used in descriptive summaries and statistical analyses, some of which may also be used for subgroup analyses. Additional covariates and other strata of clinical interest may also be considered.

| Category | Details |
|---|---|
| Strata | Age Group at Screening (5-7 years old, 8-11 years old), Ease of Use Questionnaire (Version A, Version B) |
| Covariates | Country |

### **5.4.2.** Examination of Subgroups

The list of subgroups may be used in descriptive summaries and statistical analyses. Additional subgroups of clinical interest may also be considered.

- If the percentage of subjects is small within a particular subgroup, then the subgroup categories may be refined prior to unblinding the trial.
- If the category cannot be refined further, then descriptive rather than statistical comparisons may be performed for the particular subgroup.

| Subgroup | Categories |
|---|---|
| Country | United States, Canada |
| Gender | Female, Male |
| Duration of Asthma | < 1 year, >=1 year to < 3 years, >=3 years to < 5 years, >=5 years |
| Main Current Asthma Therapy | Rescue Only, Maintenance with or without Rescue |
| Main Current Asthma Therapy | DPI, MDI, Other |
| Device Type | |

# 5.5. Multiple Comparisons and Multiplicity

There are no planned adjustments for multiple comparisons or multiplicity.

# 5.6. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:

| Section | Component |
|---------|----------------------------------------------------------------|
| 10.3 | Appendix 3: Assessment Windows |
| 10.4 | Appendix 4: Study Phases and Treatment Emergent Adverse Events |
| 10.5 | Appendix 5: Data Display Standards & Handling Conventions |
| 10.6 | Appendix 6: Derived and Transformed Data |

| Section | Component |
|---------|-----------------------------------------------------|
| 10.7 | Appendix 7: Reporting Standards for Missing Data |
| 10.8 | Appendix 8: Values of Potential Clinical Importance |

#### 6. STUDY POPULATION ANALYSES

# 6.1. Overview of Planned Study Population Analyses

The study population analyses will be based on the Intent-to-Treat (ITT) population, unless otherwise specified.

Study population analyses including analyses of participant's disposition, protocol deviations, demographic and baseline characteristics, prior and concomitant medications, and exposure and treatment compliance will be based on GSK Core Data Standards.

Details of the planned displays are presented in Appendix 10: List of Data Displays

## **6.2.** Participant Disposition

The study population summary will use the ASE population and show the number of participants overall who were screened, the number of screen failures and the number with each reason for the screen failure. The display will also showcase the number of participants who are in the ITT population (complete screening and demonstrate correct use at visit 1) and MITT population (attend visit 2 and are randomised to a version of the ease of use questionnaire).

For the ITT population, reasons for withdrawal summary will present the number and percentage of participants who completed the study, those who withdrew prematurely from the study and those who reported a primary and sub-reason for the withdrawal.

#### 6.3. Medical Conditions

The number and percentage of participants reporting each current medical condition will be presented. All medical conditions will be summarised in the displays regardless of the frequencies. This applies to both the current and past medical condition displays.

#### 6.4. Concomitant Medications

Concomitant medications will be coded using the GSK Drug coding dictionary. A summary of the number and percentage of subjects with concomitant medications will be displayed by GSK-Drug Anatomical Therapeutic Chemical (ATC) classification level 1 (Body System) and ingredient. This summary will present drugs that are composed of a combination of ingredients and will be displayed according to the ATC classifications of the ingredients (combination) and will also include single-ingredient medications. Summaries will be split into those taken pre-treatment, during treatment, and post-treatment.

#### 6.5. Incorrect Use at Visit 1

Participants will be asked to demonstrate correct use of the ELLIPTA at visit 1. The participants will have up to 5 attempts to demonstrate correct use. The number of participants who attempt correct use will be presented along with the number and percentages of those who did not demonstrate correct use after attempts number 1 to 5. The number and percentages of each item not performed correctly at each attempt will be summarised in the display for all participants. The summary will be based on the ITT population.

#### 7. EFFICACY ANALYSES

## 7.1. Primary Efficacy Analyses

The primary analyses will include:

- To determine the proportion of participants from each stratum who demonstrate correct use of the ELLIPTA DPI after the study period at V2.
- To determine the proportion of participants from each stratum who rate the use of the ELLIPTA DPI as easy to use, from those who could demonstrate correct use of the ELLIPTA DPI after the study period at V2.

#### 7.1.1. Endpoints

The primary endpoints are:

- The percentage of participants from each stratum who demonstrate correct use of the ELLIPTA DPI after the study period at V2.
- The percentage of participants from each stratum who rate the ELLIPTA DPI as easy to use, from those who could demonstrate correct use of the ELLIPTA DPI after the study period at V2.

## 7.1.2. Summary Measure

The percentage for both endpoints will be reported for each stratum for the single treatment group along with a 95% confidence interval (CI) for the percentage, calculated using the exact binomial distribution.

## 7.1.3. Population of Interest

The primary efficacy analyses will be based on the Modified Intent-to-Treat (MITT) population, unless otherwise specified.

## 7.1.4. Strategy for Intercurrent (Post-Randomization) Events

The MITT population composes of participants who have been screened, received at least one dose of the study medication (placebo) and were randomized to a version of the ease of use questionnaire at V2. Therefore, we can only identify intercurrent events that occur at V2 only.

Intercurrent events are defined as:

- Early discontinuation of study drug
- Early withdrawal from study (not completing correct use checklist or ease of use questionnaire)
- Use of prohibited medications

The "Treatment policy" strategy will be applied to handle the "Use of prohibited medications" and "Early discontinuation of drug" in the analysis for all endpoints. The strategy implies direct use of data irrespective of the occurrence of the intercurrent

events. This means the participant's data will be included in the analysis regardless whether they discontinued the ELLIPTA DPI placebo or used a prohibited medication at Visit 2. The "Treatment policy" strategy is the same as de facto type estimand. The strategy for the Early withdrawal from study intercurrent events is mentioned below for the endpoints.

# 7.1.4.1. Percentage of participants from each stratum who demonstrate correct use of the ELLIPTA DPI after the study period at V2.

The "Composite" strategy will be used for the "Early withdrawal from study" intercurrent event. Participants who make it to V2 will be randomised to a version of the ease of use questionnaire and complete this questionnaire. The participants will then be asked to demonstrate correct use of the ELLIPTA DPI. A participant is expected to complete the full demonstration, however there is a possibility the participant might choose to no longer participate and not complete the full demonstration (i.e. decide to stop half way through the demonstration of the required steps for correct use of the ELLIPTA DPI). In the occurrence of this intercurrent event, the endpoint will be the percentage of participants from each stratum who demonstrate correct use of the ELLIPTA DPI after the study period at V2, where those who are deemed "not correct use" will comprise of the participants who did not demonstrate correct use of the ELLIPTA DPI and those who did not complete the demonstration of correct use. The strategy modifies the definition of the summary measure, such that the intercurrent event becomes a component of the outcome. A footnote will be included on displays to indicate this composite endpoint, if this intercurrent event should occur.

If a participant withdraws from the study, or a parent no longer consents their child before the correct use demonstration can be started, then they will be deemed an early withdrawal and no data will be collected for this endpoint.

# 7.1.4.2. Percentage of participants from each stratum who rate the ELLIPTA DPI as easy to use, from those who could demonstrate correct use of the ELLIPTA DPI after the study period at V2.

The "Composite" strategy will be used for the "Early withdrawal from study" intercurrent event. Participants who make it to V2 will be randomised to a version of the ease of use questionnaire, asked to complete the questionnaire and then will perform a demonstration of correct use of the ELLIPTA DPI. The first question relates to the ease of use of the ELLIPTA DPI, while the second question relates to the ease of telling the number of doses remaining in the ELLIPTA DPI. A participant is expected to complete the questionnaire before the correct use demonstration, however there is a possibility the participant might only answer one or zero of the questions, and still able to perform the correct use demonstration, or choose to no longer participate in the study. In the occurrence of this intercurrent event, the endpoint will be the percentage of participants from each stratum who rate the ELLIPTA DPI as easy to use, from those who could demonstrate correct use of the ELLIPTA DPI after the study period at V2, where those who rate the ease of use of ELLIPTA DPI as "hard" comprise of the participants who rated the ELLIPTA DPI as "hard" and those who did not answer the ease of use question. A footnote will be included on displays to indicate this composite endpoint, if this intercurrent event should occur.

If a participant withdraws from the study, or a parent no longer consents their child before the questionnaire can be started, then they will be deemed an early withdrawal and no data will be collected for this endpoint.

#### 7.1.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 10: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 7.1.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed

#### 7.1.5.1. Statistical Methodology Specification

# 7.1.5.1.1. Percentage of participants from each stratum who demonstrate correct use of the ELLIPTA DPI after the study period at V2

#### **Endpoint / Variables**

• The percentage of participants from each stratum who demonstrate correct use of the ELLIPTA DPI after the study period at V2.

#### **Model Specification**

- The primary endpoint of the percentage of participants from each stratum who demonstrate correct use of the ELLIPTA DPI after the study period at V2 will be analysed using the Modified Intent-to-Treat population.
  - This endpoint will be analysed using the exact binomial distribution to calculate the 95% CI

#### **Model Checking & Diagnostics**

 Computation of the confidence intervals for the proportions is based on the exact (Clopper-Pearson) binomial distribution.

#### **Model Results Presentation**

 The percentage will be reported for each stratum for the single treatment group along with a 95% confidence interval (CI) for the percentage, calculated using the exact binomial distribution.

#### **Sensitivity and Supportive Analyses**

 Observed analyses: Along with the primary composite estimand display, an observed data display with no imputation may be presented if a substantial amount (10% of the total population) of participants do not complete the correct use demonstration. This display will include the correct use demonstration completers only.

# 7.1.5.1.2. Percentage of participants from each stratum who rate the ELLIPTA DPI as easy to use, from those who could demonstrate correct use of the ELLIPTA DPI after the study period at V2

#### **Endpoint / Variables**

 The percentage of participants from each stratum who rate the ELLIPTA DPI as easy to use, from those who could demonstrate correct use of the ELLIPTA DPI after the study period at V2.

#### **Model Specification**

- The primary endpoint of the percentage of participants from each stratum who rate the ELLIPTA DPI as easy to use, from those who could demonstrate correct use of the ELLIPTA DPI after the study period at V2 will be analysed using the Modified Intent-to-Treat population.
  - This endpoint will be analysed using the exact binomial distribution to calculate the 95% CI

#### **Model Checking & Diagnostics**

Computation of the confidence intervals for the proportions is based on the exact (Clopper-Pearson) binomial distribution.

#### **Model Results Presentation**

 The percentage will be reported for each stratum for the single treatment group along with a 95% confidence interval (CI) for the percentage, calculated using the exact binomial distribution.

### Sensitivity and Supportive Analyses

 Observed analyses: Along with the primary composite estimand display, an observed data display with no imputation may be presented if a substantial amount (10% of the total population) of participants do not answer ease of use questionnaire. This display will include the ease of use question completers only.

# 7.2. Secondary Efficacy Analyses

The secondary efficacy analyses will include:

- To determine the proportion of participants from each stratum who demonstrate correct use of the ELLIPTA DPI after initial training from HCP only at V1.
- To determine the proportion of participants who demonstrate correct use of the ELLIPTA DPI after the study period at V2.
- To determine the proportion of participants who rate the use of the ELLIPTA DPI as easy to use, from those who could demonstrate correct use of the ELLIPTA DPI after the study period at V2.
- To determine the proportion of participants from each stratum who made at least one critical error during use of the ELLIPTA DPI after initial training from HCP only at V1.

#### 7.2.1. Endpoints

The secondary endpoints are:

- The percentage of participants from each stratum who demonstrate correct use of the ELLIPTA DPI after initial training from HCP at V1.
- The percentage of participants who demonstrate correct use of the ELLIPTA DPI after the study period at V2.
- The percentage of participants who rate the ELLIPTA DPI as easy to use, from those who could demonstrate correct use of the ELLIPTA DPI after the study period at V2.
- The percentage of participants from each stratum who made at least one critical error during use of the ELLIPTA DPI after initial training from HCP at V1.

## 7.2.2. Summary Measure

The percentage for all secondary endpoints will be reported for the single treatment group along with a 95% confidence interval (CI) for the percentage, calculated using the exact binomial distribution.

#### 7.2.3. Population of Interest

The secondary efficacy analyses will be based on the Intent-To-Treat or Modified Intent-to-Treat populations, unless otherwise specified.

## 7.2.4. Strategy for Intercurrent (Post-Randomization) Events

Intercurrent events are defined as:

- Early discontinuation of study drug
- Early withdrawal from study
- Use of prohibited medications

The "Treatment policy" strategy will be applied to handle the "Use of prohibited medications" and "Early discontinuation of study drug" in the analysis for all endpoints. The strategy implies direct use of data irrespective of the occurrence of the intercurrent events. The "Treatment policy" strategy is the same as de facto type estimand. The strategy for the Early withdrawal from study intercurrent events is mentioned below for the endpoints.

# 7.2.4.1. Percentage of participants from each stratum who demonstrate correct use of the ELLIPTA DPI after initial training from HCP at V1.

The population of interest will be based on the Intent-to-Treat population.

The "Composite" strategy will be used for the "Early withdrawal from study" intercurrent event. Participants who pass the screening visit (Visit 0) will then be taught by the HCP how to correctly use the ELLIPTA DPI. The participant is then provided with their own ELLIPTA DPI and will be asked to demonstrate correct use. If the participant demonstrates correct use of the ELLIPTA DPI, they will progress through the study and

deemed correct use at V1, attempt one. If the participant cannot perform correct use on their first attempt, then they will have four more attempts, and will be deemed a "not correct use" on the first attempt. A participant is expected to complete the full correct use demonstration, however there is a possibility the participant might choose to no longer participate and not complete the full demonstration. In the occurrence of this intercurrent event, the endpoint will be the percentage of participants from each stratum who demonstrate correct use of the ELLIPTA DPI after initial training from the HCP at V1, where those who are deemed "not correct use" will comprise of participants who did not perform correct use of the ELLIPTA DPI on attempt one <u>and</u> those who did not complete the demonstration of correct use on attempt one. A footnote will be included on displays to indicate this composite endpoint, if this intercurrent event should occur.

If a participant withdraws from the study, or a parent no longer consents their child before the correct use demonstration can be started, then they will be deemed a screen failure and no data will be collected for this endpoint.

# 7.2.4.2. Percentage of participants who demonstrate correct use of the ELLIPTA DPI after the study period at V2.

The population of interest will be based on the Modified Intent-to-Treat population.

The "Composite" strategy will be used for the "Early withdrawal from study" intercurrent event. Participants who make it to V2 will be randomised to a version of the ease of use questionnaire and asked to complete the questionnaire. The participants will then be asked to demonstrate correct use of the ELLIPTA DPI. A participant is expected to complete the full demonstration, however there is a possibility the participant might choose to no longer participate and not complete the full demonstration (i.e. decide to stop half way through the demonstration of the required steps for correct use of the ELLIPTA DPI). In the occurrence of this intercurrent event, the endpoint will be the percentage of participants who demonstrate correct use of the ELLIPTA DPI after the study period at V2, where those who are deemed "not correct use" will comprise of the participants who did not demonstrate correct use of the ELLIPTA DPI and those who did not complete the demonstration of correct use. A footnote will be included on displays to indicate this composite endpoint, if this intercurrent event should occur.

If a participant withdraws from the study, or a parent no longer consents their child before the correct use demonstration can be started, then they will be deemed an early withdrawal and no data will be collected for this endpoint.

# 7.2.4.3. Percentage of participants who rate the ELLIPTA DPI as easy to use, from those who could demonstrate correct use of the ELLIPTA DPI after the study period at V2.

The population of interest will be based on the Modified Intent-to-Treat population.

The "Composite" strategy will be used for the "Early withdrawal from study" intercurrent event. Participants who make it to V2 will be randomised to a version of the ease of use questionnaire, asked to complete the questionnaire and then will perform a demonstration of correct use of the ELLIPTA DPI. The first question relates to the ease of use of the

ELLIPTA DPI, while the second question relates to the ease of telling the number of doses remaining in the ELLIPTA DPI. A participant is expected to complete the questionnaire before the correct use demonstration, however there is a possibility the participant might only answer one or zero of the questions, and still able to perform the correct use demonstration, or choose to no longer participate in the study. In the occurrence of this intercurrent event, the endpoint will be the percentage of participants who rate the ELLIPTA DPI as easy to use, from those who could demonstrate correct use of the ELLIPTA DPI after the study period at V2, where those who rate the ease of use of ELLIPTA DPI as "hard" comprise of the participants who rated the ELLIPTA DPI as "hard" and those who did not answer the ease of use question. A footnote will be included on displays to indicate this composite endpoint, if this intercurrent event should occur.

If a participant withdraws from the study, or a parent no longer consents their child before the questionnaire can be started, then they will be deemed an early withdrawal and no data will be collected for this endpoint.

# 7.2.4.4. Percentage of participants from each stratum who made at least one critical error during use of the ELLIPTA DPI after initial training from HCP at V1

The population of interest will be based on the Intent-to-Treat population.

The "Composite" strategy will be used for the "Early withdrawal from study" intercurrent event. Participants who pass the screening visit (Visit 0) will then be taught by the HCP how to correctly use the ELLIPTA DPI. The participant is then provided with their own ELLIPTA DPI and will be asked to demonstrate correct use. Four of the ten correct use checklist items are deemed as "critical errors" (see Section 10.6.3 for the details on critical errors). A participant is expected to perform throughout the whole correct use demonstration, however there is a possibility the participant might choose to no longer participate and not complete the full demonstration (i.e. only perform 2 of the 4 critical error items during the correct use demonstration). In the occurrence of this intercurrent event, the endpoint will be the percentage of participants from each stratum who made at least one critical error during use of the ELLIPTA DPI after initial training from HCP at V1. If a participant withdraws at any point throughout the correct use demonstration and performed a critical error, then the participant will be deemed as one who performed at least one critical error. If the participant withdraws at any point throughout the correct use demonstration and did not perform all the critical error items, then taking the conservative approach, the participant will also be deemed as one who performed at least one critical error. If the participant withdraws at any point during the correct use demonstration and performs all critical error items correctly, then the participant will be deemed as one who did not perform at least one critical error. A footnote will be included on displays to indicate this composite endpoint, if this intercurrent event should occur.

If a participant withdraws from the study, or a parent no longer consents their child before the correct use demonstration can be started, then they will be deemed a screen failure and no data will be collected for this endpoint.

#### 7.2.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 10: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 7.2.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

#### 7.2.5.1. Statistical Methodology Specification

# 7.2.5.1.1. Percentage of participants from each stratum who demonstrate correct use of the ELLIPTA DPI after initial training from HCP at V1

#### **Endpoint / Variables**

• The percentage of participants from each stratum who demonstrate correct use of the ELLIPTA DPI after initial training from HCP at V1.

#### **Model Specification**

- The endpoint of the percentage of participants from each stratum who demonstrate correct use
  of the ELLIPTA DPI after initial training from HCP at V1 will be analysed using the Intent-toTreat population.
  - This endpoint will be analysed using the exact binomial distribution to calculate the 95% CI

#### **Model Results Presentation**

 The percentage will be reported for each stratum for the single treatment group along with a 95% confidence interval (CI) for the percentage, calculated using the exact binomial distribution.

#### **Sensitivity and Supportive Analyses**

Observed analyses: Along with the composite estimand display, an observed data display with
no imputation may be presented if a substantial amount (10% of the total population) of
participants do not complete the correct use demonstration. This display will include the correct
use demonstration completers only.

# 7.2.5.1.2. Percentage of participants who demonstrate correct use of the ELLIPTA DPI after the study period at V2.

#### **Endpoint / Variables**

 The percentage of participants who demonstrate correct use of the ELLIPTA DPI after the study period at V2.

#### **Model Specification**

- The endpoint of the percentage of participants who demonstrate correct use of the ELLIPTA
   DPI after the study period at V2 will be analysed using the Modified Intent-to-Treat population.
  - This endpoint will be analysed using the exact binomial distribution to calculate the 95% CI

#### Model Results Presentation

• The percentage will be reported for the single treatment group along with a 95% confidence interval (CI) for the percentage, calculated using the exact binomial distribution.

### **Sensitivity and Supportive Analyses**

Observed analyses: Along with the composite estimand display, an observed data display with
no imputation may be presented if a substantial amount (10% of the total population) of
participants do not complete the correct use demonstration. This display will include the correct
use demonstration completers only.

# 7.2.5.1.3. Percentage of participants who rate the use of the ELLIPTA DPI as easy to use, from those who could demonstrate correct use of the ELLIPTA DPI after the study period at V2.

#### **Endpoint / Variables**

• The percentage of participants who rate the ELLIPTA DPI as easy to use, from those who could demonstrate correct use of the ELLIPTA DPI after the study period at V2.

#### **Model Specification**

- The endpoint of the percentage of participants who rate the ELLIPTA DPI as easy to use, from those who could demonstrate correct use of the ELLIPTA DPI after the study period at V2 will be analysed using the Modified Intent-to-Treat population.
  - This endpoint will be analysed using the exact binomial distribution to calculate the 95% CI

#### **Model Results Presentation**

• The percentage will be reported for the single treatment group along with a 95% confidence interval (CI) for the percentage, calculated using the exact binomial distribution.

#### **Sensitivity and Supportive Analyses**

 Observed analyses: Along with the primary composite estimand display, an observed data display with no imputation may be presented if a substantial amount (10% of the total population) of participants do not answer ease of use questionnaire. This display will include the ease of use question completers only.

# 7.2.5.1.4. Percentage of participants from each stratum who made at least one critical error during use of the ELLIPTA DPI after initial training from HCP at V1.

#### **Endpoint / Variables**

 The percentage of participants from each stratum who made at least one critical error during use of the ELLIPTA DPI after initial training from HCP at V1.

#### **Model Specification**

 The endpoint of the percentage of participants from each stratum who made at least one critical error during use of the ELLIPTA DPI after initial training from HCP at V1 will be analysed using the Intent-to-Treat population.

 This endpoint will be analysed using the exact binomial distribution to calculate the 95% CI

#### **Model Results Presentation**

 The percentage will be reported for each stratum for the single treatment group along with a 95% confidence interval (CI) for the percentage, calculated using the exact binomial distribution.

## **Sensitivity and Supportive Analyses**

Observed analyses: Along with the composite estimand display, an observed data display with
no imputation may be presented if a substantial amount (10% of the total population) of
participants do not complete the correct use demonstration. This display will include the correct
use demonstration completers only.

## 7.3. Exploratory Efficacy Analyses

The exploratory efficacy analyses will include:

- To determine the proportion of participants from each stratum who rate the ability to tell how many puffs are left in the ELLIPTA DPI as easy after the study period at V2.
- To determine the proportion of participant's parents/guardians who rate the ability to tell how many doses are remaining in the ELLIPTA DPI as easy or very easy after the study period at V2.
- To determine the proportion of participant's parents/guardians who would be 'likely' or 'very likely' to ask their doctor for the ELLIPTA DPI if the participants current daily inhaled medication(s) were available in the ELLIPTA DPI after the study period at V2.
- To determine the proportion of participants from each stratum who can demonstrate correct use after the study period at V2 with assistance from parents/guardians.
- To determine the proportion of participants from each stratum who made at least one critical error during use of the ELLIPTA DPI after the study period at V2.
- To determine the proportion of participants who made at least one critical error during use of the ELLIPTA DPI after initial training from HCP at V1.

## 7.3.1. Endpoints

The exploratory efficacy endpoints are:

- The percentage of participants from each stratum who rate the ability to tell how many puffs are left in the ELLIPTA DPI as easy after the study period at V2.
- The percentage of participant's parents/guardians who rate the ability to tell how many doses are remaining in the ELLIPTA DPI as easy or very easy after the study period at V2.

- The percentage of participant's parents/guardians who would be likely or very likely to ask their doctor for the ELLIPTA DPI if the participants current daily inhaled medication(s) were available in the ELLIPTA DPI after the study period at V2.
- The percentage of participants from each stratum who demonstrated correct use after the study period at V2 with assistance from parents/guardians.
- The percentage of participants from each stratum who made at least one critical error during use of the ELLIPTA DPI after the study period at V2.
- The percentage of participants who made at least one critical error during use of the ELLIPTA DPI after initial training from HCP at V1.

### 7.3.2. Summary Measures

The percentage for all exploratory efficacy endpoints will be reported for the single treatment group along with a 95% confidence interval (CI) for the percentage, calculated using the exact binomial distribution.

### 7.3.3. Population of Interest

The exploratory efficacy analyses will be based on the Intent-To-Treat or Modified Intent-to-Treat populations, unless otherwise specified.

### 7.3.4. Strategy for Intercurrent (Post-Randomization) Events

Intercurrent events are defined as:

- Early discontinuation of study drug
- Early withdrawal from study
- Use of prohibited medications

The "Treatment policy" strategy will be applied to handle the "Use of prohibited medications" and "Early discontinuation of study drug" in the analysis for all endpoints. The strategy implies direct use of data irrespective of the occurrence of the intercurrent events. The "Treatment policy" strategy is the same as de facto type estimand. The strategy for the Early withdrawal from study intercurrent events is mentioned below for the endpoints.

# 7.3.4.1. Percentage of participants from each stratum who rate the ability to tell how many puffs are left in the ELLIPTA DPI as easy after the study period at V2

The population of interest will be based on the Modified Intent-to-Treat population.

The "Composite" strategy will be used for the "Early withdrawal from study" intercurrent event. Participants who make it to V2 will be randomised to a version of the ease of use questionnaire, asked to complete the questionnaire and then will perform a demonstration of correct use of the ELLIPTA DPI. The first question relates to the ease of use of the ELLIPTA DPI, while the second question relates to the ease of telling the number of doses remaining in the ELLIPTA DPI. A participant is expected to complete the questionnaire before the correct use demonstration, however there is a possibility the

participant might only answer one or zero of the questions, and still able to perform the correct use demonstration, or choose to no longer participate in the study. In the occurrence of this intercurrent event, the endpoint will be the percentage of participants who rate the ability to tell how many puffs are left in the ELLIPTA DPI as easy after the study period at V2, where those who rate the ease of telling the number of puffs remaining in the ELLIPTA DPI as "hard" comprise of the participants who answered the question as "hard" and those who did not answer the ease of number of puffs question. A footnote will be included on displays to indicate this composite endpoint, if this intercurrent event should occur.

If a participant withdraws from the study, or a parent no longer consents their child before the questionnaire can be started, then they will be deemed an early withdrawal and no data will be collected for this endpoint.

# 7.3.4.2. Percentage of participant's parents/guardians who rate the ability to tell how many doses are remaining in the ELLIPTA DPI as easy or very easy after the study period at V2.

The population of interest will be based on the Modified Intent-to-Treat population.

The "Composite" strategy will be used for the "Early withdrawal from study" intercurrent event. Participants who make it to V2 will be randomised to a version of the ease of use questionnaire and asked to complete the questionnaire. The parent/guardian will also be given the same version (A or B) of their own questionnaire. The parent's questionnaire contains two questions, and these relate to: the ease or difficulty of telling how many doses were left in the ELLIPTA DPI, and whether you would be likely to request your child's asthma medication in the ELLIPTA DPI if it were available. Similarly, as the participant, the parent is expected to fully complete the questionnaire, however there is a possibility the parent might only answer one or zero of the questions or choose to no longer allow their child to participate in the study. In the occurrence of this intercurrent event, the endpoint will be the percentage of participant's parents/guardians who rate the ability to tell how many doses are remaining in the ELLIPTA DPI as easy or very easy after the study period at V2, where those who rate the ease of telling the number of doses remaining in the ELLIPTA DPI other than "easy" or "very easy" comprise of the participants parents who answered the question as "hard" or "very hard" and those who did not answer the ease of number of doses question. These parents will be grouped as "Hard/Very Hard" i.e. those parents who do not answer the question will contribute to the overall denominator of the population. A footnote will be included on displays to indicate this composite endpoint, if this intercurrent event should occur.

If a participant withdraws from the study, or a parent no longer consents their child before the questionnaire can be started, then they will be deemed an early withdrawal and no data will be collected for this endpoint.

# 7.3.4.3. Percentage of participant's parents/guardians who would be likely or very likely to ask their doctor for the ELLIPTA DPI if the participants current daily inhaled medication(s) were available in the ELLIPTA DPI after the study period at V2.

The population of interest will be based on the Modified Intent-to-Treat population.

The "Composite" strategy will be used for the "Early withdrawal from study" intercurrent event. This endpoint will use the same strategy as detailed in 7.3.4.2. In the occurrence of this intercurrent event, the endpoint will be the percentage of participant's parents/guardians who would be likely or very likely to ask their doctor for the ELLIPTA DPI if the participants current daily inhaled medication(s) were available in the ELLIPTA DPI after the study period at V2, where those who answer the second question of the ease of use questionnaire other than "likely" or "very likely" comprise of the participants parents who answered the question as "unlikely" or "very unlikely" <a href="mailto:and-those who did not answer the second ease of use question.">and those who did not answer the second ease of use question. These parents will be grouped as "Unlikely/Very Unlikely". i.e. those parents who do not answer the question will contribute to the overall denominator of the population. A footnote will be included on displays to indicate this composite endpoint, if this intercurrent event should occur.

If a participant withdraws from the study, or a parent no longer consents their child before the questionnaire can be started, then they will be deemed an early withdrawal and no data will be collected for this endpoint.

# 7.3.4.4. Percentage of participants from each stratum who demonstrate correct use after the study period at V2 with assistance from parents/guardians

The population of interest will be based on the Modified Intent-to-Treat population.

The "Composite" strategy will be used for the "Early withdrawal from study" intercurrent event. Participants who make it to V2 will be randomised to a version of the ease of use questionnaire, asked to complete the questionnaire and then will perform a demonstration of correct use of the ELLIPTA DPI. After a participant has performed the demonstration of correct use, they will either have performed it correctly and finish the study or have not demonstrated correct use and will be asked to try again with the assistance of their parent/guardian. A similar strategy will be applied for this intercurrent event as detailed in 7.1.4.1. In the occurrence of this intercurrent event, the endpoint will be the percentage of participants from each stratum who demonstrate correct use of the ELLIPTA DPI after the study period at V2 with assistance from parents/guardians, where those who are deemed "not correct use" will comprise of the participants who did not demonstrate correct use of the ELLIPTA DPI and those who did not complete the demonstration of correct use. A footnote will be included on displays to indicate this composite endpoint, if this intercurrent event should occur.

If a participant withdraws from the study, or a parent no longer consents their child before the correct use demonstration can be started, then they will be deemed an early withdrawal and no data will be collected for this endpoint.

# 7.3.4.5. Percentage of participants from each stratum who made at least one critical error during use of the ELLIPTA DPI after the study period at V2.

The population of interest will be based on the Modified Intent-to-Treat population.

The "Composite" strategy will be used for the "Early withdrawal from study" intercurrent event. This endpoint only considers the first correct use attempt at visit 2, and not both correct use attempts (i.e. the second attempt with the assistance from the parent/guardian is not included). A similar strategy for this incurrent event will be applied as detailed in 7.2.4.4. In the occurrence of this intercurrent event, the endpoint will be the percentage of participants from each stratum who made at least one critical error during use of the ELLIPTA DPI after the study period at V2. If a participant withdraws at any point throughout the correct use demonstration and performed a critical error, then the participant will be deemed as one who performed at least one critical error. If the participant withdraws at any point throughout the correct use demonstration and did not perform all the critical error items, then taking the conservative approach, the participant will also be deemed as one who performed at least one critical error. If the participant withdraws at any point during the correct use demonstration and performs all critical error items correctly, then the participant will be deemed as one who did not perform at least one critical error. A footnote will be included on displays to indicate this composite endpoint, if this intercurrent event should occur.

If a participant withdraws from the study, or a parent no longer consents their child before the correct use demonstration can be started, then they will be deemed an early withdrawal and no data will be collected for this endpoint.

# 7.3.4.6. Percentage of participants who made at least one critical error during use of the ELLIPTA DPI after initial training from HCP at V1.

The population of interest will be based on the Intent-to-Treat population.

The "Composite" strategy will be used for the "Early withdrawal from study" intercurrent event. A similar strategy for this incurrent event will be applied as detailed in 7.2.4.4. In the occurrence of this intercurrent event, the endpoint will be the percentage of participants who made at least one critical error during use of the ELLIPTA DPI after initial training from HCP at V1. If a participant withdraws at any point throughout the correct use demonstration and performed a critical error, then the participant withdraws at any point throughout the correct use demonstration and did not perform all the critical error items, then taking the conservative approach, the participant will also be deemed as one who performed at least one critical error. If the participant withdraws at any point during the correct use demonstration and performs all critical error items correctly, then the participant will be deemed as one who did not perform at least one critical error. A footnote will be included on displays to indicate this composite endpoint, if this intercurrent event should occur.

If a participant withdraws from the study, or a parent no longer consents their child before the correct use demonstration can be started, then they will be deemed a screen failure and no data will be collected for this endpoint.

### 7.3.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 10: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 7.3.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed

#### 7.3.5.1. Statistical Methodology Specification

7.3.5.1.1. Percentage of participants from each stratum who rate the ability to tell how many puffs are left in the ELLIPTA DPI as easy after the study period at V2

#### **Endpoint / Variables**

• The percentage of participants from each stratum who rate the ability to tell how many puffs are left in the ELLIPTA DPI as easy after the study period at V2

### **Model Specification**

- The endpoint of the percentage of participants from each stratum who rate the ability to tell
  how many puffs are left in the ELLIPTA DPI as easy after the study period at V2 will be
  analysed using the Modified Intent-to-Treat population.
  - This endpoint will be analysed using the exact binomial distribution to calculate the 95% CI

#### **Model Results Presentation**

• The percentage will be reported for the single treatment group along with a 95% confidence interval (CI) for the percentage, calculated using the exact binomial distribution.

#### **Sensitivity and Supportive Analyses**

 Observed analyses: Along with the primary composite estimand display, an observed data display with no imputation may be presented if a substantial amount (10% of the total population) of participants do not answer ease of use questionnaire. This display will include the number of puffs question completers only.

# 7.3.5.1.2. Percentage of participant's parents/guardians who rate the ability to tell how many doses are remaining in the ELLIPTA DPI as easy or very easy after the study period at V2.

#### **Endpoint / Variables**

The percentage of participants parents/guardians who rate the ability to tell how many doses
are remaining in the ELLIPTA DPI as easy or very easy after the study period at V2.

#### **Model Specification**

- The endpoint of the percentage of participants parents/guardians who rate the ability to tell
  how many doses are remaining in the ELLIPTA DPI as easy or very easy after the study period
  at V2 will be analysed using the Modified Intent-to-Treat population.
  - This endpoint will be analysed using the exact binomial distribution to calculate the 95% CI

#### **Model Results Presentation**

• The percentage will be reported for the single treatment group along with a 95% confidence interval (CI) for the percentage, calculated using the exact binomial distribution.

#### Sensitivity and Supportive Analyses

- Observed analyses: Along with the primary composite estimand display, an observed data display with no imputation may be presented if a substantial amount (10% of the total population) of participants parents/guardians do not answer ease of use questionnaire. This display will include the number of doses question completers only.
- It is required for the parent/guardian who attends visit 2 to have also attended visit 1. A
  sensitivity analysis may be presented if a substantial amount (10% of the total population) of
  participants parents/guardians who attend visit 2 are not the same as those who attended visit
  1. This display will only include the results of those parents/guardians who attended both study
  visits.
- 7.3.5.1.3. Percentage of participant's parents/guardians who would be likely or very likely to ask their doctor for the ELLIPTA DPI if the participants current daily inhaled medication(s) were available in the ELLIPTA DPI after the study period at V2.

#### **Endpoint / Variables**

 The percentage of participant's parents/guardians who would be likely or very likely to ask their doctor for the ELLIPTA DPI if the participants current daily inhaled medication(s) were available in the ELLIPTA DPI after the study period at V2.

#### **Model Specification**

The endpoint of the participant's parents/guardians who would be likely or very likely to ask
their doctor for the ELLIPTA DPI if the participants current daily inhaled medication(s) were
available in the ELLIPTA DPI after the study period at V2 will be analysed using the Modified

Intent-to-Treat population.

 This endpoint will be analysed using the exact binomial distribution to calculate the 95% CI

#### **Model Results Presentation**

• The percentage will be reported for the single treatment group along with a 95% confidence interval (CI) for the percentage, calculated using the exact binomial distribution.

#### **Sensitivity and Supportive Analyses**

- Observed analyses: Along with the primary composite estimand display, an observed data display with no imputation may be presented if a substantial amount (10% of the total population) of participants parents/guardians do not answer ease of use questionnaire. This display will include the current daily inhaled medication question completers only.
- It is required for the parent/guardian who attends visit 2 to have also attended visit 1. A sensitivity analysis may be presented if a substantial amount (10% of the total population) of participants parents/guardians who attend visit 2 are not the same as those who attended visit 1. This display will only include the results of those parents/guardians who attended both study visits.

# 7.3.5.1.4. Percentage of participants from each stratum who demonstrate correct use after the study period at V2 with assistance from parents/guardians

#### **Endpoint / Variables**

• The percentage of participants from each stratum who demonstrate correct use after the study period at V2 with assistance from parents/guardians.

#### **Model Specification**

- The endpoint of the participants from each stratum who demonstrate correct use after the study period at V2 with assistance from parents/guardians will be analysed using the Modified Intent-to-Treat population.
  - This endpoint will be analysed using the exact binomial distribution to calculate the 95% CI

#### **Model Results Presentation**

• The percentage will be reported for the single treatment group along with a 95% confidence interval (CI) for the percentage, calculated using the exact binomial distribution.

#### Sensitivity and Supportive Analyses

- Observed analyses: Along with the composite estimand display, an observed data display with
  no imputation may be presented if a substantial amount (10% of the total population) of
  participants do not complete the correct use demonstration. This display will include the correct
  use demonstration completers only.
- It is required for the parent/guardian who attends visit 2 to have also attended visit 1. A sensitivity analysis may be presented if a substantial amount (10% of the total population) of participants parents/guardians who attend visit 2 are not the same as those who attended visit

1. This display will only include the results of those parents/guardians who attended both study visits.

# 7.3.5.1.5. Percentage of participants from each stratum who made at least one critical error during use of the ELLIPTA DPI after the study period at V2.

#### **Endpoint / Variables**

• The percentage of participants from each stratum who made at least one critical error during use of the ELLIPTA DPI after the study period at V2.

#### **Model Specification**

- The endpoint of the participants from each stratum who made at least one critical error during use of the ELLIPTA DPI after the study period at V2 will be analysed using the Modified Intentto-Treat population.
  - This endpoint will be analysed using the exact binomial distribution to calculate the 95% CI

#### Model Results Presentation

• The percentage will be reported for the single treatment group along with a 95% confidence interval (CI) for the percentage, calculated using the exact binomial distribution.

#### **Sensitivity and Supportive Analyses**

Observed analyses: Along with the composite estimand display, an observed data display with
no imputation may be presented if a substantial amount (10% of the total population) of
participants do not complete the correct use demonstration. This display will include the correct
use demonstration completers only.

# 7.3.5.1.6. Percentage of participants who made at least one critical error during use of the ELLIPTA DPI after initial training from HCP at V1.

#### **Endpoint / Variables**

 The percentage of participants who made at least one critical error during use of the ELLIPTA DPI after initial training from HCP at V1.

#### **Model Specification**

- The endpoint of the participants who made at least one critical error during use of the ELLIPTA DPI after initial training from HCP at V1 will be analysed using the Modified Intent-to-Treat population.
  - This endpoint will be analysed using the exact binomial distribution to calculate the 95% CI

#### **Model Results Presentation**

The percentage will be reported for the single treatment group along with a 95% confidence

interval (CI) for the percentage, calculated using the exact binomial distribution.

### **Sensitivity and Supportive Analyses**

Observed analyses: Along with the composite estimand display, an observed data display with
no imputation may be presented if a substantial amount (10% of the total population) of
participants do not complete the correct use demonstration. This display will include the correct
use demonstration completers only.

#### 8. SAFETY ANALYSES

The safety analyses will be based on the ITT population, unless otherwise specified.

#### 8.1. Adverse Events

Adverse events analyses including summaries of adverse events (AEs), serious adverse events (SAEs) and any other significant AE's will be based on the GSK Core Data Standards.

Considering this is a placebo only ELLIPTA DPI study and no active drug is being prescribed, the summaries will be presented for all participants combined regardless of their randomised questionnaire version. The details of the planned analyses are provided in Appendix 10: List of Data Displays

A summary of the following AEs and SAEs will be provided:

- Any AE or SAE (pre-treatment (SAE only), on-treatment or post-treatment)]
- Any on-treatment drug related AE
- Any on-treatment non-serious AE
- Any AE (pre-treatment or on-treatment) leading to permanent discontinuation of study treatment or withdrawal from the study
- Any fatal AE
- Any non-fatal SAE
- Any on-treatment non-fatal drug related SAE
- Any on-treatment fatal drug related SAE

The numbers and percentage of participants will all AEs (regardless of causality) will be summarised by system organ class (SOC) and preferred term (PT). The ordering of the SOCs and PTs will be in descending order of total incidence. A SOC will not be presented if the overall incidence for AE within the particular system. If the total incidence for any two or more AEs is equal, the events will be presented in alphabetical order

# 8.2. Adverse Events of Special Interest Analyses

No AE of special interest analysis will be performed as no active drug is prescribed in this study.
# 9. REFERENCES

GlaxoSmithKline Document Number 2017N346371\_00 Study ID 206924. An open-label study to evaluate correct use and ease of use of the ELLIPTA Dry Powder Inhaler (DPI) in pediatric patients currently receiving inhaled therapy for treatment of their asthma. Report Date 23-Jan-2018.

# 10. APPENDICES

# 10.1. Appendix 1: Protocol Deviation Management

The full list of protocol deviations collected on the eCRF is in the Protocol Deviation Management Plan (PDMP). Please refer to this document for current guidance.

# 10.1.1. Exclusions from Per Protocol Population

There is no Per Protocol population in this study.

# 10.2. Appendix 2: Schedule of Activities

# 10.2.1. Protocol Defined Schedule of Events

| | Visit 0- | Tre | eatment Per | iod | |
|---|---|---|---|---|---|
| Procedure | Screeni<br>ng<br>(up to<br>30 days<br>before<br>Day 1) | Visit 1<br>(can<br>occur on<br>same day<br>as<br>screenin<br>g) | Early<br>Withdra<br>wal | Visit 2 | Notes |
| Study Day | -30 | 1 | | 29 ± 2 | All assessments concern study participants only, unless otherwise stated (parent/guardians). |
| Screening | | | | | |
| Informed consent and assent | Х | | | | Visit 1 must occur within 30 days of signing of providing informed consent. Must be signed before any study procedures. Assent must be provided. |
| Inclusion and exclusion criteria | Х | | | | All of the inclusion and none of the exclusion criteria must be met prior to inclusion at V0. This includes ability to demonstrate correct use of the ELLIPTA DPI after training. |
| Demography | Х | | | | Age, sex, race, ethnicity. |
| Physical Examination | Х | | | | Including height and weight, |
| Concomitant medications | Х | | | | Concomitant medications pertaining to the participant's diagnosis of asthma collected (minimum previous 3 months). |
| Past and current medical conditions | Х | | | | |
| Asthma History | Х | | | | Participant will have a medical history of symptoms consistent with a diagnosis of asthma. |
| Exacerbation History | Х | | | | Asthma exacerbation history for the previous year will be collected. |
| Randomization | | | | Х | Randomization refers to the version of the questionnaire only. |
| Safety | | | | | |
| AE review | | ←===== | ======= | <del>-</del> | Collected from Visit 1 until the completion of the final assessment at Visit 2. |
| SAE review | <b>←====</b> | | | | Collected from time of informed consent/assent until the completion of the final assessment at Visit 2. |
| Concomitant medications review | <b>←====</b> | ======= | ======= | <del>-</del> | Review any changes in concomitant medications. |
| Asthma exacerbations | <b>←====</b> | <del>-</del> | | | Asthma exacerbation information will be collected for the duration of the study (see Section 9.2.6 in the Protocol). |
| Questionnaires and Asses | ssments | | | | |
| First training in correct use of ELLIPTA DPI by HCP | | Х | | | Initial training by HCP |
| Correct use of ELLIPTA DPI after first instruction by HCP | | Х | | | First demonstration of correct use of ELLIPTA DPI. |

| | Visit 0- | Tre | Treatment Period | | |
|---|---|---|---|---|---|
| Procedure | Screeni<br>ng<br>(up to<br>30 days<br>before<br>Day 1) | Visit 1<br>(can<br>occur on<br>same day<br>as<br>screenin<br>g) | Early<br>Withdra<br>wal | Visit 2 | Notes |
| Second and third training in correct use of ELLIPTA DPI by HCP | | X | | | Training only if necessary (participant made errors) |
| Correct use of ELLIPTA DPI<br>after second and third<br>instruction by HCP | | Х | | | Second and third demonstrations of correct use of ELLIPTA DPI |
| Fourth and fifth training in correct use of ELLIPTA DPI by HCP and parent/guardian | | Х | | | Training only if necessary (participant made errors) |
| Correct use of ELLIPTA DPI after fourth and fifth instruction by HCP and parent/guardian | | X | | | Fourth and fifth demonstrations of correct use of ELLIPTA DPI. After which time they will be registered as a screen failure if correct use has not been demonstrated. |
| Ease of use Questionnaire completion | | | | Х | This is completed upon return to the site after the study period. This must occur before any other assessments at V2. |
| Compliance with ELLIPTA DPI | | | Х | Х | This will be taken from the dose counter. |
| Correct use of ELLIPTA DPI after treatment period | | | | Х | Demonstration of correct use of ELLIPTA DPI without any instruction at V2. |
| Correct use of ELLIPTA DPI with instruction from parent/guardian | | | | Х | Demonstration of correct use of ELLIPTA DPI with instruction from parent/guardian at V2. Only necessary if correct use is not demonstrated during first attempt. |
| Placebo ELLIPTA DPI | | | | | |
| Dispense Placebo ELLIPTA DPI(s) | | Х | | | Procedures for dispensation and return of clinical supplies will be described in detail in the Study Reference Manual (SRM). If a participant |
| Return Placebo ELLIPTA DPI | | X | Х | Х | completes all study requirements, they will need 2 ELLIPTA DPIs. One will remain at site and the other will be used during the study period. |

AE – Adverse Event, DPI - Dry Powder Inhaler, HCP - Healthcare Professional, SAE - Serious Adverse Events,

# 10.3. Appendix 3: Assessment Windows

# 10.3.1. Definitions of Assessment Windows for Analyses

Study day  $29 \pm 2$  (Visit 2, 28 days after Visit 1) is defined as the day of randomisation to an ease of use questionnaire.

| Analysis Set | Parameter | Target | Analysis | Analysis | |
|---|---|---|---|---|---|
| / Domain | (if applicable) | | Beginning<br>Timepoint | Ending<br>Timepoint | Timepoint |
| | All | 1 | -30 | 1 | Visit 0 |
| | All | 1 | 1 | 1 | Visit 1 |
| | All | 29 | 27 | 31 | Visit 2 |

#### NOTES:

• Visit 1 can occur on same day as screening visit (Visit 0)

# 10.4. Appendix 4: Study Phases and Treatment Emergent Adverse Events

# 10.4.1. Study Phases

Assessments and events will be classified according to the time of occurrence relative to study treatment start and stop dates.

| Study Phase | Definition |
|---|---|
| Pre-Treatment | Date < Study Treatment Start Date |
| On-Treatment | Study Treatment Start Date ≤ Date ≤ Study Treatment Stop Date + 1 |
| Post-Treatment | Date > Study Treatment Stop Date + 1 |

# 10.4.1.1. Study Phases for Concomitant Medication

Treatment phases for summaries of Asthma and Non-Asthma concomitant medications will be defined as follows:

| Definition | Treatment Phase | | |
|---|---|---|---|
| Delinition | Pre-Treatment | On-Treatment | Post-Treatment |
| Subject did not take study treatment (e.g, screening failures) and conmed stop date > date of Screening or variable that asks if conmed is on-going (refer hereafter as ongoingmed) is "yes" | Υ | | |
| (Conmed start date < treatment start date or variable that asks if medication taken prior to study is "yes"(refer hereafter as priormed)) and date of Screening < conmed stop date < treatment start date | Υ | | |
| (Conmed start date < treatment start date or priormed is yes) and (treatment start date ≤ conmed stop date ≤ treatment stop date) | Y | Y | |
| (Conmed start date < treatment start date or priormed is yes) and (conmed stop date > treatment stop date or ongoingmed is "yes") | Y | Y | Υ |
| (Treatment start date ≤ conmed start date < treatment stop date and treatment start date ≤ conmed stop date ≤ treatment stop date) or (Treatment start date = conmed start date = conmed stop date) | | Y | |
| (Treatment start date ≤ conmed start date < treatment stop date) or (Treatment start date = conmed start date = treatment stop date) and (conmed stop date > treatment stop date or ongoingmed is Yes) | | Y | Υ |

| Definition | Treatment Phase | | |
|---|---|---|---|
| Delillition | Pre-Treatment | On-Treatment | Post-Treatment |
| Conmed start ≥ treatment stop date and | | | Y |
| treatment start date ≠ treatment stop date | | | l |

#### NOTES:

- A concomitant medication will be classed in every period of the study in which it was taken (e.g., run-in, on-treatment or post-treatment).
- See Section 10.7.2.1 for handling of partial dates.
- If the study treatment stop date is missing, it will be imputed as described in Section 10.7.
- Medications that stopped prior to Screening will not be assigned a treatment phase and will not be summarized.

# 10.4.2. Treatment Emergent Flag for Adverse Events

| Flag | Definition |
|---|---|
| Treatment | If AE onset date is on or after Visit 1 start date & on or before Visit 2 stop date. |
| Emergent | <ul> <li>(Visit 1 Start Date ≤ AE Start Date ≤ Visit 2 Stop Date + 1 day).</li> </ul> |

#### NOTES:

If the study treatment stop date is missing, then the AE will be considered to be On-Treatment.

# 10.5. Appendix 5: Data Display Standards & Handling Conventions

### 10.5.1. Reporting Process

| Software | |
|---|---|
| The currently supported versions of SAS software will be used. | |
| Reporting Area | |
| HARP Server | : UK1SALX00175 |
| HARP Compound | : GSK2285997 |
| QC Spreadsheet | : gsk2285997/mid206924/final_01/documents |
| Analysis Datasets | |
| <ul> <li>Analysis datasets will be created according to CDISC standards (SDTM IG Version 3.2 &amp; ADaM IG<br/>Version 1.0.</li> </ul> | |
| Generation of RTF Files | |
| RTF files will be | RTF files will be generated for use in writing the CSR. |

### 10.5.2. Reporting Standards

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated (IDSL Standards Location: https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics
- Do not include subject level listings in the main body of the GSK Clinical Study Report. All subject level listings should be located in the modular appendices as ICH or non-ICH listings

#### **Formats**

- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF.

### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days
    on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.

#### **Unscheduled Visits**

- Unscheduled visits will not be included in summary tables and/or figures.
- All unscheduled visits will be included in listings.

| Descriptive Summary Statistics | |
|---|---|
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | N, n, frequency, % |
| Graphical Displays | |
| Refer to IDSL Statistical Principals 7.01 to 7.13. | |

### 10.6. Appendix 6: Derived and Transformed Data

#### 10.6.1. General

#### **Study Day**

- Calculated as the number of days from First Dose Date:
  - Ref Date = Missing → Study Day = Missing
  - Ref Date < First Dose Date → Study Day = Ref Date First Dose Date</li>
  - Ref Data ≥ First Dose Date → Study Day = Ref Date (First Dose Date) + 1

### 10.6.2. Study Population

#### **Treatment Compliance**

For ELLIPTA inhaler, the number of doses of study inhaler taken by each subject will be calculated from the dose counter start and stop counts for each inhaler prescribed during the 4-week study period (take home period). The derivation for treatment compliance during the 4-week study period is defined as the sum of (Dose Counter Start-Dose Counter Stop) over all inhalers dispensed to the participant and returned during the 4-week study period. If a dose counter start count is missing, then it will be assumed to be 30. If dose counter stop count is non-missing, then the percentage compliance will be calculated as:

$$Compliance = \frac{(\textit{Total Number of Inhalations Taken})}{(\textit{Treatment Stop Date} - \textit{Treatment Start Date} + 1)} \times 100$$

Where **Total Number of Inhalations Taken** is the total number of doses taken from all ELLIPTA DPI placebo inhalers in the 4-week study period, and **Treatment Start Date** and **Treatment Stop Date** are the earliest treatment start date and the latest treatment stop date recorded for all of the inhalers used in the calculation.

 If the dose counter stop count is missing for the subject, then the treatment compliance will be set to missing for that subject.

#### **Extent of Exposure**

Number of days of exposure to study drug will be calculated based on the formula:

#### Duration of Exposure in Days = Treatment Stop Date - (Treatment Start Date) + 1

- Participants who successfully complete the Visit 1 assessments but did not report a treatment start date will be categorised as having zero days of exposure.
- If there are any treatment breaks during the study, exposure data will be adjusted accordingly.

#### 10.6.3. **Efficacy**

#### **Correct Use Checklist**

#### **Demonstrate Correct Use**

For a participant to have demonstrated correct use, they need to have a "Yes" to all the correct use checklist items recorded:

- Participant slides the cover completely down to expose the mouthpiece until a "click" is heard.
- Participant does not shake the inhaler
- Participant breathes out (exhales) while holding the inhaler away from their mouth
- Participant does not breathe into the mouthpiece
- Participant places mouthpiece between lips, and closes lips firmly around it.
- Participant takes one long steady deep breath in through their mouth

#### **Correct Use Checklist**

- Participant does not block air vent with fingers.
- Participant removes inhaler from his/her mouth and holds his/her breath
- Participant breathes out slowly and gently
- Participant closes the inhaler completely

#### **Critical Errors**

If a participant has recorded a "No" to any of the following in the correct use checklist items, this is then considered a critical error for the ELLIPTA DPI:

- Participant slides the cover completely down to expose the mouthpiece until a "click" is heard.
- Participant does not shake the inhaler
- Participant does not breathe into the mouthpiece
- Participant places mouthpiece between lips, and closes lips firmly around it.

#### **Ease of Use Questionnaire**

#### **Number of Doses Remaining**

The number of participant's parents/guardians who answer the number of doses question in their respective versions of the questionnaire as "Easy" or "Very easy" will be summarised together and presented such as:

- Very easy
- Easy
- Difficult
- Very difficult
- Very easy/Easy

The 95% confident intervals will be calculated for all the responses listed above using the exact binomial distribution.

#### **Current Inhaled Asthma Medication**

The number of participant's parents/guardians who answer the current inhaled asthma medication question in their respective versions of the questionnaire as "Likely" or "Very likely" will be summarised together and presented such as:

- Very likely
- Likely
- Unlikely
- Very unlikely
- Very likely/Likely

The 95% confident intervals will be calculated for all the responses listed above using the exact binomial distribution.

### 10.6.4. Safety

Safety is only summarised in this study – no derivations or transformations are required.

# 10.7. Appendix 7: Reporting Standards for Missing Data

# 10.7.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Subject study completion (i.e. as specified in the protocol) was defined as one who has completed all phases of the study (Visit 0 through Visit 2).</li> <li>Withdrawn subjects will not be replaced in the study.</li> </ul> |
| | All available data from participants who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified. |
| | Withdrawal visits will be slotted as per Appendix 3: Assessment Windows or will be summarised as withdrawal visits. |

# 10.7.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: |
| | <ul> <li>These data will be indicated by the use of a "blank" in subject listing displays.</li> <li>Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> </ul> |
| | <ul> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be<br/>missing data and should be displayed as such.</li> </ul> |
| Outliers | Any participants excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

# 10.7.2.1. Handling of Missing and Partial Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |
| Adverse<br>Events | <ul> <li>The eCRF allows for the possibility of partial dates (i.e., only month and year) to be recorded for AE start and end dates; that is, the day of the month may be missing. In such a case, the following conventions will be applied for calculating the time to onset and the duration of the event: <ul> <li>Missing Start Day: First of the month will be used unless this is before the start date of study treatment; in this case the study treatment start date will be used and hence the event is considered On-treatment as per Appendix 4: Study Phases and Treatment Emergent Adverse Events.</li> <li>Missing Stop Day: Last day of the month will be used, unless this is after the stop date of study treatment; in this case the study treatment stop date will be used.</li> </ul> </li> <li>Completely missing start or end dates will remain missing, with no imputation applied.</li> <li>Start or end dates which are completely missing (i.e. no year specified) will remain missing, with no imputation applied.</li> </ul> |
| Concomitant<br>Medications/<br>Medical<br>History | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention:</li> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month.</li> </ul> |

| Element | Reporting Detail |
|---|---|
| | <ul> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent<br/>on the month and year) and 'Dec' will be used for the month.</li> </ul> |
| | The recorded partial date will be displayed in listings. |

# 10.8. Appendix 8: Values of Potential Clinical Importance

# 10.8.1. Vital Signs

Height, weight, gestational age and gestational weight will be collected and presented in this study.

As this is a placebo only ELLIPTA DPI study, there are no values of potential clinical importance.

# 10.9. Appendix 9: Abbreviations & Trade Marks

# 10.9.1. Abbreviations

| Abbreviation | Description |
|--------------|------------------------------------------------|
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| ASE | All Subjects Enrolled |
| A&R | Analysis and Reporting |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| CS | Clinical Statistics |
| CSR | Clinical Study Report |
| DBF | Database Freeze |
| DBR | Database Release |
| DOB | Date of Birth |
| DP | Decimal Places |
| DPI | Dry Powder Inhaler |
| eCRF | Electronic Case Record Form |
| GSK | GlaxoSmithKline |
| ICF | Informed Consent Form |
| ICH | International Conference on Harmonization |
| IDMC | Independent Data Monitoring Committee |
| IDSL | Integrated Data Standards Library |
| IMMS | International Modules Management System |
| IP | Investigational Product |
| ITT | Intent-To-Treat |
| MITT | Modified Intent-to-Treat |
| PDMP | Protocol Deviation Management Plan |
| QC | Quality Control |
| RAP | Reporting & Analysis Plan |
| RAMOS | Randomization & Medication Ordering System |
| SAC | Statistical Analysis Complete |
| SDTM | Study Data Tabulation Model |
| SOP | Standard Operation Procedure |
| TA | Therapeutic Area |
| TFL | Tables, Figures & Listings |

# 10.9.2. Trademarks

| Trademarks of the GlaxoSmithKline<br>Group of Companies |
|---------------------------------------------------------|
| ELLIPTA |

| Trademarks not owned by the GlaxoSmithKline Group of Companies | |
|----------------------------------------------------------------|---|
| SAS | • |

# 10.10. Appendix 10: List of Data Displays

# 10.10.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------|-------------------|------------|
| Study Population | 1.1 to 1.29 | N/A |
| Efficacy | 2.1 to 2.16 | 2.1 to 2.4 |
| Safety | 3.1 to 3.16 N/A | |
| Section | List | ings |
| ICH Listings | Listings 1 to 20 | |
| Other Listings | Listings 21 to 32 | |

### 10.10.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required example mock-up displays provided in Appendix 11: Example Mock Shells for Data Displays

| Section | Figure | Table | Listing |
|------------------|--------|---------|---------|
| Study Population | N/A | POP_Tn | POP_Ln |
| Efficacy | EFF_Fn | EFF_Tn | EFF_Ln |
| Safety | N/A | SAFE_Tn | SAFE_Ln |

#### NOTES:

Non-Standard displays are indicated in the 'IDSL / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

#### 10.10.3. Deliverables

| Delivery [Priority] [1] | Description |
|-------------------------|-------------------------------------|
| Dry Run [1] | Dry Run Deliverable before DBR |
| SAC [2] | Final Statistical Analysis Complete |

#### NOTES:

<sup>1.</sup> Indicates priority (i.e. order) in which displays will be generated for the reporting effort

# 10.10.4. Study Population Tables

| Study F | Population Tabl | les | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subject | Disposition | | | | • |
| 1.1. | ASE | SP1 | Summary of Study Populations | Present by 5-7 year, 8-11 year, Total columns | Dry Run[1]<br>SAC[2] |
| 1.2. | ASE | ES6 | Summary of Screening Status and Reasons for Screen Failure | Present by 5-7 year, 8-11 year, Total columns | Dry Run[1]<br>SAC[2] |
| 1.3. | ASE | NS1 | Summary of Number of Participants by Country and Site ID | Present by 5-7 year, 8-11 year, Total columns | Dry Run[1]<br>SAC[2] |
| 1.4. | ITT | Non-standard<br>POP_T1 | Summary of Attendance at Each Clinical Visit | Present by 5-7 year, 8-11 year, Total columns | Dry Run[1]<br>SAC[2] |
| 1.5. | ITT | SD1 | Summary of Treatment Status and Reasons for Discontinuation of Study Treatment | Present by 5-7 year, 8-11 year, Total columns | Dry Run[1]<br>SAC[2] |
| 1.6. | ITT | ES1 | Summary of End of Study Record | Present by 5-7 year, 8-11 year, Total columns | Dry Run[1]<br>SAC[2] |
| 1.7. | ITT | ES4 | Summary of Participant Disposition at Each Epoch | Present by 5-7 year, 8-11 year, Total columns | Dry Run[1]<br>SAC[2] |
| Protoco | ol Deviations | | | | |
| 1.8. | ASE | DV1 | Summary of Important Protocol Deviations – All Subjects<br>Enrolled Population | Present by 5-7 year, 8-11 year, Total columns | Dry Run[1]<br>SAC[2] |
| 1.9. | ASE | IE1 | Summary of Inclusion/Exclusion/Randomisation Criteria Deviations – All Subjects Enrolled Population | Present by 5-7 year, 8-11 year, Total columns | Dry Run[1]<br>SAC[2] |
| 1.10. | ITT | DV1 | Summary of Important Protocol Deviations – Intent-to-Treat Population | Present by 5-7 year, 8-11 year, Total columns | Dry Run[1]<br>SAC[2] |

| Study I | Population Tab | les | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.11. | ITT | IE1 | Summary of Inclusion/Exclusion/Randomisation Criteria Deviations - Intent-to-Treat Population | Present by 5-7 year, 8-11 year, Total columns | Dry Run[1]<br>SAC[2] |
| Popula | tion Analysed | | | | |
| 1.12. | ITT | SP2 | Summary of Exclusions from the Modified Intent-to-Treat Population | Present by 5-7 year, 8-11 year, Total columns | Dry Run[1]<br>SAC[2] |
| Demog | raphic and Bas | eline Characteris | tics | | |
| 1.13. | ITT | DM1 | Summary of Demographic Characteristics | Present by 5-7 year, 8-11 year, Total columns | Dry Run[1]<br>SAC[2] |
| 1.14. | ASE | DM11 | Summary of Age Ranges | Present Total Column only | Dry Run[1]<br>SAC[2] |
| 1.15. | ITT | DM5 | Summary of Race and Racial Combinations | Present Total Column only | Dry Run[1]<br>SAC[2] |
| 1.16. | ITT | DM6 | Summary of Race and Racial Combinations Details | Present Total Column only | Dry Run[1]<br>SAC[2] |
| 1.17. | ITT | Non-standard<br>POP_T5 | Summary of Subgroups | Present by 5-7 year, 8-11 year, Total columns | Dry Run[1]<br>SAC[2] |
| Medica | Medical Conditions & Concomitant Medications | | | | |
| 1.18. | ITT | MH4 | Summary of Current Medical Conditions | Present Total Column only | Dry Run[1]<br>SAC[2] |
| 1.19. | ITT | MH4 | Summary of Past Medical Conditions | Present Total Column only | Dry Run[1]<br>SAC[2] |

| Study F | Population Tab | les | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.20. | ITT | Non-standard<br>POP_T2 | Summary of Duration of Asthma and Asthma Exacerbation History at Screening | Present Total Column only | Dry Run[1]<br>SAC[2] |
| 1.21. | ITT | CM1 | Summary of Pre-Treatment Asthma Concomitant Medications | Present 5-7 year, 8-11 year, Total columns | Dry Run[1]<br>SAC[2] |
| 1.22. | ITT | CM1 | Summary of Pre-Treatment Non-Asthma Concomitant Medications | Present 5-7 year, 8-11 year, Total columns | Dry Run[1]<br>SAC[2] |
| 1.23. | ITT | CM1 | Summary of On-Treatment Asthma Concomitant Medications | Present 5-7 year, 8-11 year, Total columns | Dry Run[1]<br>SAC[2] |
| 1.24. | ITT | CM1 | Summary of On-Treatment Non-Asthma Concomitant Medications | Present 5-7 year, 8-11 year, Total columns | Dry Run[1]<br>SAC[2] |
| 1.25. | ITT | CM1 | Summary of Post-Treatment Asthma Concomitant Medications | Present 5-7 year, 8-11 year, Total columns | Dry Run[1]<br>SAC[2] |
| 1.26. | ITT | CM1 | Summary of Post-Treatment Non-Asthma Concomitant Medications | Present 5-7 year, 8-11 year, Total columns | Dry Run[1]<br>SAC[2] |
| Exposi | re and Treatmo | ent Compliance | | | |
| 1.27. | ITT | Non-standard<br>POP_T3 | Summary of Exposure to Study Treatment | Present 5-7 year, 8-11 year, Total columns | Dry Run[1]<br>SAC[2] |
| 1.28. | ITT | Non-standard<br>POP_T4 | Summary of Study Compliance | Present 5-7 year, 8-11 year, Total columns | Dry Run[1]<br>SAC[2] |

| Study P | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Summa | ry of Intercurre | ent Events | | | |
| 1.29. | ITT | Non-standard<br>POP_T6 | Summary of Intercurrent Events | Present 5-7 year, 8-11 year, Total columns | Dry Run[1]<br>SAC[2] |

# 10.10.5. Efficacy Tables

| Efficac | y: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Correct | Use | | | | |
| 2.1. | ITT | EFF_T1 | Summary of the Number of Completers of the Correct Use Demonstration at Visit 1 | | Dry Run [1]<br>SAC [2] |
| 2.2. | ASE | EFF_T11 | Summary of Number of Attempts to Demonstrate Correct Use of ELLIPTA at Visit 1 – All Subjects Enrolled | Present 5-7 year, 8-11 year, Total columns Note: Attempts 1, 2 and 3 the Healthcare Professional trains the participant in correct use of the ELLIPTA DPI. Attempts 4 and 5 the parents/guardians assist the participant in demonstrating correct use of the ELLIPTA DPI. Programming Note: Percentages are based on the subjects who attempted to demonstrate correct use, not Big N. | Dry Run [1]<br>SAC [2] |
| 2.3. | ITT | EFF_T11 | Summary of Number of Attempts to Demonstrate Correct Use of ELLIPTA at Visit 1 – Intent-to-Treat Population | Present 5-7 year, 8-11 year, Total columns Note: Attempts 1, 2 and 3 the Healthcare Professional trains the participant in correct use of the ELLIPTA DPI. Attempts 4 and 5 the parents/guardians assist the participant in demonstrating correct use of the ELLIPTA DPI. Programming Note: Percentages are based on the subjects who attempted to demonstrate correct use, not Big N. | Dry Run [1]<br>SAC [2] |

| Efficacy | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.4. | ITT | EFF_T2 | Summary of Correct Use at Visit 1 | Repeat for attempts 2 to 5. | Dry Run[1]<br>SAC [2] |
| 2.5. | ITT | EFF_T10 | Summary of Critical Errors at Visit 1 | Repeat for attempts 2 to 5. | Dry Run[1]<br>SAC [2] |
| 2.6. | MITT | EFF_T1 | Summary of the Number of Completers of the Correct Use Demonstration at Visit 2 | | Dry Run [1]<br>SAC [2] |
| 2.7. | MITT | EFF_T2 | Summary of Correct Use at Visit 2 | Repeat for attempt 2 | Dry Run [1]<br>SAC [2] |
| 2.8. | ITT | EFF_T10 | Summary of Critical Errors at Visit 2 | Repeat for attempt 2 | Dry Run [1]<br>SAC [2] |
| 2.9. | MITT | EFF_T11 | Summary of Number of Attempts to Demonstrate Correct Use of ELLIPTA at Visit 2 | Present 5-7 year, 8-11 year, Total columns Programming Note: Only include Number of Attempts: 1, 2 or Did not perform correct use after 2 attempts. Note: Attempt 1 the participant attempts to demonstrate correct use of the ELLIPTA DPI. Attempt 2 the parents/guardians assist the participant in demonstrating correct use of the ELLIPTA DPI. Programming Note: Percentages are based on the subjects who attempted to demonstrate correct use, not Big N. | Dry Run [1]<br>SAC [2] |
| Ease of | Use at Visit 2 | | | | |
| 2.10. | MITT | EFF_T9 | Summary of the Number of Completers of the Ease of Use Questionnaire at Visit 2 | | Dry Run [1]<br>SAC [2] |

| Efficacy | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.11. | MITT | EFF_T3 | Summary of Participants Ease of Use at Visit 2 | Present by: "Questionnaire: Overall, Version A, Version B" | Dry Run [1]<br>SAC [2] |
| 2.12. | MITT | EFF_T4 | Summary of Parent/Guardians Ease of Use at Visit 2 | Present by: "Questionnaire: Overall, Version A, Version B" | Dry Run [1]<br>SAC [2] |
| Protoco | ol Defined Endp | oints for Correct | Use and Ease of Use | | • |
| 2.13. | MITT | EFF_T5 | Summary of Protocol Defined Endpoints for Correct Use and Ease of Use at Visit 2 by Age Stratum | | Dry Run [1]<br>SAC [2] |
| 2.14. | MITT | EFF_T6 | Summary of Protocol Defined Endpoints for Correct Use and Ease of Use at Visit 2 | | Dry Run [1]<br>SAC [2] |
| 2.15. | ITT | EFF_T7 | Summary of Protocol Defined Endpoints for Correct Use at End of Visit 1 by Age Stratum | | Dry Run [1]<br>SAC [2] |
| 2.16. | ITT | EFF_T8 | Summary of Protocol Defined Endpoints for Correct Use at End of Visit 1 | | Dry Run [1]<br>SAC [2] |

# 10.10.6. Efficacy Figures

| Efficacy | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Correct | Use | | | | |
| 2.1. | ITT | EFF_F1 | Summary of Correct Use at Visit 1 | Present Age Stratum: 5-7 Year Old, 8-11 Year Old on one page, and Total Population on the second page Note: Attempts 1, 2 and 3 the Healthcare Professional trains the participant in correct use of the ELLIPTA DPI. Attempts 4 and 5 the parents/guardians assist the participant in demonstrating correct use of the ELLIPTA DPI. | Dry Run [1]<br>SAC [2] |
| 2.2. | MITT | EFF_F1 | Summary of Correct Use at Visit 2 | Present Age Stratum: 5-7 Year Old, 8-11 Year Old on one page, and Total Population on the second page Present only Attempts "Overall", "1" and "2" Note: Attempt 1 the participant attempts to demonstrate correct use of the ELLIPTA DPI. Attempt 2 the parents/guardians assist the participant in demonstrating correct use of the ELLIPTA DPI. | Dry Run [1]<br>SAC [2] |

| Efficacy | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.3. | MITT | EFF_F2 | Summary of Participant's Ease of Use at Visit 2 | Present Age Stratum: 5-7 Year Old, 8- 11 Year Old on one page, and Total Population on the second page Replace "Number of Doses" and "Request the ELLIPTA" with "Ease of Use" and Number of Puffs". Include footnotes: Ease of Use: Responder is defined as the number of participants who rate the use of ELLIPTA as easy Number of Puffs: Responder is defined as the number of participants who rate the ability to tell how many doses are remaining in the ELLIPTA as easy | Dry Run [1]<br>SAC [2] |
| 2.4. | MITT | EFF_F2 | Summary of Parent/Guardian's Ease of Use at Visit 2 | Present Age Stratum: 5-7 Year Old, 8-<br>11 Year Old on one page, and Total<br>Population on the second page. | Dry Run [1]<br>SAC [2] |

# 10.10.7. Safety Tables

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | e Events | | | | |
| 3.1. | ITT | AE13 | Adverse Event Overview | Present Total column only Note: All participants received placebo only ELLIPTA DPI Inhalers. | Dry Run [1]<br>SAC [2] |
| 3.2. | ITT | AE1 | Summary of Adverse Events by System Organ Class and Preferred Term | Present Total column only Note: All participants received placebo only ELLIPTA DPI Inhalers. | Dry Run [1]<br>SAC [2] |
| 3.3. | ITT | AE1 | Summary of On-Treatment Adverse Events by System Organ Class and Preferred Term | Present Total column only Note: All participants received placebo only ELLIPTA DPI Inhalers. | Dry Run [1]<br>SAC [2] |
| 3.4. | ITT | AE1 | Summary of Drug-Related Adverse Events | Present Total column only Note: All participants received placebo only ELLIPTA DPI Inhalers. | Dry Run [1]<br>SAC [2] |
| 3.5. | ITT | AE1 | Summary of Non-Serious Drug Related Adverse Events | Present Total column only Note: All participants received placebo only ELLIPTA DPI Inhalers. | Dry Run [1]<br>SAC [2] |
| 3.6. | ITT | AE3 | Summary of Common (>=3%) Adverse Events by Overall Frequency | Present Total column only Note: All participants received placebo only ELLIPTA DPI Inhalers. | Dry Run [1]<br>SAC [2] |
| 3.7. | ITT | AE15 | Summary of Common (>=3%) On-Treatment Non-Serious<br>Adverse Events by Overall Frequency (Number of Subjects and<br>Occurrences) | Present Total column only Note: All participants received placebo only ELLIPTA DPI Inhalers. | Dry Run [1]<br>SAC [2] |
| 3.8. | ITT | AE15 | Summary of Common (>=3%) Non-Serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | Present Total column only Note: All participants received placebo only ELLIPTA DPI Inhalers. | Dry Run [1]<br>SAC [2] |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.9. | ITT | AE15 | Summary of Common (>=3%) On-Treatment Drug Related Adverse Events by Overall Frequency (Number of Subjects and Occurrences) | Present Total column only Note: All participants received placebo only ELLIPTA DPI Inhalers. | Dry Run [1]<br>SAC [2] |
| 3.10. | ASE | AE16 | Summary of Serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | Present Total column only Note: All participants received placebo only ELLIPTA DPI Inhalers. | Dry Run [1]<br>SAC [2] |
| 3.11. | ITT | AE16 | Summary of On-Treatment Serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | Present Total column only Note: All participants received placebo only ELLIPTA DPI Inhalers. | Dry Run [1]<br>SAC [2] |
| 3.12. | ITT | AE1 | Summary of Serious Drug Related Adverse Events | Present Total column only Note: All participants received placebo only ELLIPTA DPI Inhalers. | Dry Run [1]<br>SAC [2] |
| 3.13. | ITT | AE1 | Summary of On-Treatment Adverse Events Leading to<br>Permanent Discontinuation of Study Drug or Withdrawal<br>from the Study | Present Total column only Note: All participants received placebo only ELLIPTA DPI Inhalers. | Dry Run [1]<br>SAC [2] |
| 3.14. | ITT | AE15 | Summary of Common (>=3%) On-Treatment Serious Adverse<br>Events by Overall Frequency (Number of Subjects and<br>Occurrences) | Present Total column only Note: All participants received placebo only ELLIPTA DPI Inhalers. | Dry Run [1]<br>SAC [2] |
| 3.15. | ITT | AE1 | Summary of Fatal Adverse Events | Present Total column only Note: All participants received placebo only ELLIPTA DPI Inhalers. | Dry Run [1]<br>SAC [2] |
| Exacer | bations | | | | |
| 3.16. | ITT | SAFE_T1 | Summary of On-Treatment Asthma Exacerbations | Present Total column only If more than 10 Asthma exacerbations are recorded, then present the summary, otherwise present listing only. | Dry Run [1]<br>SAC [2] |

# 10.10.8. ICH Listings

| ICH Lis | tings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Study F | Population | | | | |
| Subjec | t Disposition | | | | |
| 1. | ASE | ES7 | Listing of Reasons for Screen Failure | Programming Note: If IDSL shell includes a treatment column, replace treatment column with "Age Stratum" column. | Dry Run [1]<br>SAC [2] |
| 2. | ITT | ES2 | Listing of Reasons for Study Withdrawal | Programming Note: If IDSL shell includes a treatment column, replace treatment column with "Age Stratum" column. | Dry Run [1]<br>SAC [2] |
| 3. | ITT | SD2 | Listing of Reasons for Study Treatment Discontinuation | Programming Note: If IDSL shell includes a treatment column, replace treatment column with "Age Stratum" column. | Dry Run [1]<br>SAC [2] |
| 4. | MITT | TA1 | Listing of Planned and Actual Ease of Use Questionnaire | Programming Note: If IDSL shell includes a treatment column, replace treatment column with "Age Stratum" column. | Dry Run [1]<br>SAC [2] |
| Protoco | ol Deviations | | | | |
| 5. | ITT | DV2 | Listing of Important Protocol Deviations | Programming Note: If IDSL shell includes a treatment column, replace treatment column with "Age Stratum" column. | Dry Run [1]<br>SAC [2] |
| 6. | ITT | IE3 | Listing of Inclusion/Exclusion/Randomisation Criteria Deviations | Programming Note: If IDSL shell includes a treatment column, replace treatment column with "Age Stratum" column. | Dry Run [1]<br>SAC [2] |

| ICH Lis | tings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 7. | ASE | SP3 | Listing of Participants Excluded from the Modified Intent-to-Treat Population | Programming Note: If IDSL shell includes a treatment column, replace treatment column with "Age Stratum" column. | Dry Run [1]<br>SAC [2] |
| Demog | raphy | | | | |
| 8. | ASE | DM2 | Listing of Demographic Characteristics | Programming Note: If IDSL shell includes a treatment column, replace treatment column with "Age Stratum" column. Programming Note: Include gestational age, gestational weight and country as the optional measurements. | Dry Run [1]<br>SAC [2] |
| 9. | ITT | DM9 | Listing of Race | Programming Note: If IDSL shell includes a treatment column, replace treatment column with "Age Stratum" column. | Dry Run [1]<br>SAC [2] |
| Exposu | ıre | | | | |
| 10. | ITT | EX3 | Listing of Exposure Data | Programming Note: If IDSL shell includes a treatment column, replace treatment column with "Age Stratum" column. | Dry Run [1]<br>SAC [2] |
| Concor | mitant Medicati | ons | | | |
| 11. | ITT | CM3 | Listing of Concomitant Medications | Programming Note: If IDSL shell includes a treatment column, replace treatment column with "Age Stratum" column. Include columns: "Pre-Treatment" "On-Treatment" "Post-Treatment" | Dry Run [1]<br>SAC [2] |

| ICH Lis | ICH Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Safety | | | | | |
| Advers | e Events | | | | |
| 12. | ITT | AE8 | Listing of All Adverse Events | Programming Note: If IDSL shell includes a treatment column, replace treatment column with "Age Stratum" column. | Dry Run [1]<br>SAC [2] |
| 13. | ITT | AE7 | Listing of Subject Numbers for Individual Adverse Events | Programming Note: If IDSL shell includes a treatment column, replace treatment column with "Age Stratum" column. | Dry Run [1]<br>SAC [2] |
| 14. | ITT | AE2 | Listing of Relationship Between Adverse Event System Organ Classes, Preferred Terms, and Verbatim Text | Programming Note: If IDSL shell includes a treatment column, replace treatment column with "Age Stratum" column. | Dry Run [1]<br>SAC [2] |
| 15. | ITT | AE8 | Listing of Adverse Events Leading to Permanent Discontinuation of Study Treatment or Withdrawal from Study | Programming Note: If IDSL shell includes a treatment column, replace treatment column with "Age Stratum" column. | Dry Run [1]<br>SAC [2] |
| 16. | ITT | AE8 | Listing of All Serious Adverse Events | Programming Note: If IDSL shell includes a treatment column, replace treatment column with "Age Stratum" column. | Dry Run [1]<br>SAC [2] |
| 17. | ITT | AE8 | Listing of Fatal Serious Adverse Events | Programming Note: If IDSL shell includes a treatment column, replace treatment column with "Age Stratum" column. | Dry Run [1]<br>SAC [2] |

| ICH Lis | ICH Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 18. | ITT | AE8 | Listing of Non-Fatal Serious Adverse Events | Programming Note: If IDSL shell includes a treatment column, replace treatment column with "Age Stratum" column. | Dry Run [1]<br>SAC [2] |
| 19. | ITT | AE8 | Listing of Reasons for Considering as a Serious Adverse Event | Programming Note: If IDSL shell includes a treatment column, replace treatment column with "Age Stratum" column. | Dry Run [1]<br>SAC [2] |
| 20. | ITT | AE8 | Listing of Other Significant Adverse Events | Programming Note: If IDSL shell includes a treatment column, replace treatment column with "Age Stratum" column. | Dry Run [1]<br>SAC [2] |

# 10.10.9. Non-ICH Listings

| Non-IC | Non-ICH Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Study F | Study Population | | | | |
| Subjec | t Disposition | | | | |
| 21. | ASE | Non-Standard<br>POP_L4 | Listing of Participants by Country and Site IDs | | Dry Run [1]<br>SAC [2] |
| Compli | ance | | | | |
| 22. | ITT | Non-Standard<br>POP_L1 | Listing of Treatment Compliance | | Dry Run [1]<br>SAC [2] |
| Medica | I Conditions & | Concomitant Med | lications | | |
| 23. | ITT | MH2 | Listing of Medical Conditions | Programming Note: If IDSL shell includes a treatment column, replace treatment column with "Age Stratum" column. | Dry Run [1]<br>SAC [2] |
| 24. | ITT | CM6 | Relationship between ATC Level 1, Ingredient and Verbatim text | Programming Note: If IDSL shell includes a treatment column, replace treatment column with "Age Stratum" column. | Dry Run [1]<br>SAC [2] |
| 25. | ITT | Non-Standard<br>POP_L2 | Listing of Asthma History and Asthma Exacerbation History | | Dry Run [1]<br>SAC [2] |
| Correc | t Use at Visit 1 | | | | |
| 26. | ITT | Non-Standard<br>POP_L3 | Listing of Correct Use at Visit 1 | | Dry Run [1]<br>SAC [2] |

| Non-IC | H Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Safety | | | | | |
| Advers | e Events | | | | |
| 27. | ITT | Non-Standard<br>SAFE_L1 | Listing of Asthma Exacerbations | | Dry Run [1]<br>SAC [2] |
| 28. | ITT | Non-Standard<br>SAFE_L2 | Listing of Deaths | Programming Note: If IDSL shell includes a treatment column, replace treatment column with "Age Stratum" column. | Dry Run [1]<br>SAC [2] |
| Efficac | у | | | | |
| Correc | t Use at Visit 2 | | | | |
| 29. | MITT | Non-standard<br>EFF_L1 | Listing of Correct Use at Visit 2 | | Dry Run [1]<br>SAC [2] |
| Ease of | Use | | | | |
| 30. | MITT | Non-standard<br>EFF_L2 | Listing of Ease of Use at Visit 2 | | Dry Run [1]<br>SAC [2] |
| 31. | MITT | Non-standard<br>EFF_L2 | Listing of Parent/Guardian Ease of Use at Visit 2 | Footnote: Q1: How easy or difficult (difficult or easy) was it for you to tell how many doses were left in the ELLIPTA inhaler? Q2: If your child's current inhaled asthma medication was available in the ELLIPTA inhaler, how likely would you be to request the ELLIPTA inhaler from your child's doctor? | Dry Run [1]<br>SAC [2] |

206924

# 10.11. Appendix 11: Example Mock Shells for Data Displays

Example: POP\_T1 Page 1 of n

Protocol: 206924 Population: Intent-to-Treat

Table 1.x Summary of Attendance at Each Clinical Visit

| Visit | 5-7 Year<br>Stratum<br>(N=xxx) | 8-11 Year<br>Stratum<br>(N=xxx) | Total<br>(N=xxx) |
|---|---|---|---|
| Visit 0 Screening (Can occur on same day as V1) | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Visit 1 Assessment (Can occur on same day as V0) | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Visit 2 Last Visit/End of Study/Early Withdrawal | xxx (xx%) | xxx (xx%) | xxx (xx%) |

206924

Example: POP\_T2
Protocol: 206924

Population: Intent-to-Treat

Table 1.xx
Summary of Asthma History and Asthma Exacerbation History at Screening

| | 5-7 Year<br>Stratum<br>(N=xxx) | 8-11 Year<br>Stratum<br>(N=xxx) | Total<br>(N=xxx) |
|---|---|---|---|
| Duration of Asthma | | | |
| n | XXX | XXX | XXX |
| < 1 year | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| >= 1 year to < 3 years | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| >= 3 years to < 5 years | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| >= 5 years | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Number of exacerbations that required Oral/Systemic | | | |
| Corticosteroids and/or antibiotics in the past 12 months | | | |
| n | XXX | XXX | XXX |
| 0 | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| 1 | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| 2 | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| >2 | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Number of exacerbations that required hospitalisation in the | | | |
| past 12 months | | | |
| n | XXX | XXX | XXX |
| 0 | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| 1 | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| 2 | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| >2 | xxx (xx%) | xxx (xx%) | xxx (xx%) |

206924

Example: POP\_T3
Protocol: 206924

Population: Intent-to-Treat

Table 1.xx Summary of Exposure

| | 5-7 Year<br>Stratum<br>(N=xxx) | 8-11 Year<br>Stratum<br>(N=xxx) | Total<br>(N=xxx) |
|---|---|---|---|
| Exposure (days) | | | |
| n | XXX | XXX | XXX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. | XX | XX | XX |
| Max. | xx | XX | XX |
| Range of exposure (days) | | | |
| n | xxx | XXX | XXX |
| < 14 | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| >= 14 | xxx (xx%) | xxx (xx%) | xxx (xx%) |
206924

Example: POP\_T4
Protocol: 206924

Population: Intent-to-Treat

Table 1.xx Summary of Study Compliance

| | 5-7 Year<br>Stratum<br>(N=xxx) | 8-11 Year<br>Stratum<br>(N=xxx) | Total<br>(N=xxx) |
|---|---|---|---|
| Compliance (%) | | | |
| n | XXX | XXX | XXX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. | XX | XX | XX |
| Max. | XX | XX | XX |
| Compliance category | | | |
| n | XXX | XXX | XXX |
| <80% | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| >=80% to <95% | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| >=95% to <=105% | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| >105% to <=120% | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| >120% | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Non-calculable | xxx (xx%) | xxx (xx%) | xxx (xx%) |

Example: POP\_T5 Page 1 of n

Protocol: 206924 Population: Intent-to-Treat

Table 1.xx Summary of Subgroups

| | 5-7 Year<br>Stratum<br>(N=xxx) | Stratum Stratum | | Stratum Stratum | Stratum Stratum | Stratum Stratum | Stratum Stratum |
|---|---|---|---|---|---|---|---|
| Country | | | | | | | |
| n | XXX | XXX | XXX | | | | |
| United States | xxx (xx%) | xxx (xx%) | xxx (xx%) | | | | |
| Canada | xxx (xx%) | xxx (xx%) | xxx (xx%) | | | | |
| Main Current Asthma Therapy | | | | | | | |
| n | XXX | XXX | XXX | | | | |
| Maintenance with/without Rescue | xxx (xx%) | xxx (xx%) | xxx (xx%) | | | | |
| Rescue Only | xxx (xx%) | xxx (xx%) | xxx (xx%) | | | | |
| Main Current Asthma Therapy Device Type | | | | | | | |
| n | XXX | XXX | XXX | | | | |
| DPI | xxx (xx%) | xxx (xx%) | xxx (xx%) | | | | |
| MDI | xxx (xx%) | xxx (xx%) | xxx (xx%) | | | | |
| Other [1] | xxx (xx%) | xxx (xx%) | xxx (xx%) | | | | |

<sup>[1]</sup> Other includes 'device' types such as Nebuliser, Pill/Tablet etc.

206924

Example: POP\_T6
Protocol: 206924

Population: Intent-to-Treat

### Table 1.xx Summary of Intercurrent Events

| | 5-7 Year<br>Stratum | 8-11 Year<br>Stratum | Total |
|---|---|---|---|
| Intercurrent events, n (%) | (N=XXX) | (N=xxx) | (N=xxx) |
| Any intercurrent event | | | |
| n | XX | XX | XX |
| Participant not fully completing the correct use demonstration at Visit 1 | xx (xx%) | xx (xx%) | xx (xx%) |
| Participant not fully completing the correct use demonstration at Visit 2 | xx (xx%) | xx (xx%) | xx (xx%) |
| Participant not fully completing the ease of use questionnaire | xx (xx%) | xx (xx%) | xx (xx%) |
| Participant's parents/guardians not fully completing the ease | xx (xx%) | xx (xx%) | xx (xx%) |
| of use questionnaire | | | |
| Early discontinuation of study ELLIPTA DPI placebo during the 4 week period | xx (xx%) | xx (xx%) | xx (xx%) |
| Participant changed their standard Asthma therapy inhaler to one contained in ELLIPTA DPI | xx (xx%) | xx (xx%) | xx (xx%) |

206924

Protocol: 206924

Population: Intent-to-Treat

Table 2.1
Summary of the Number of Completers of the Correct Use Demonstration at Visit 1

| Attempt: 1 | 5-7 Year<br>Stratum<br>(N=xxx) | 8-11 Year<br>Stratum<br>(N=xxx) | Total<br>(N=xxx) |
|---|---|---|---|
| Number of participants who attempted to demonstrate correct use of the ELLIPTA DPI [1] | xxx | xxx | xxx |
| Number of participants who completed the ELLIPTA correct use demonstration [2] | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Number of participants who did not fully complete the ELLIPTA DPI correct use demonstration [3] | xxx (xx%) | xxx (xx%) | xxx (xx%) |

Note: Attempts 1, 2 and 3 the Healthcare Professional trains the participant in correct use of the ELLIPTA DPI. Attempts 4 and 5 the parents/guardians assist the participant in demonstrating correct use of the ELLIPTA DPI.

- [1] The participants who attempted to demonstrate correct use of the ELLIPTA DPI at that attempt.
- [2] The participants who completed the correct use demonstration whether they correctly demonstrated or not.
- [3] The participants who did not fully perform the correct use demonstration. These participants will be assumed to have not demonstrated correct use.

Programming Note: Repeat for Attempt: 2 to 5.

Example: EFF\_T2
Protocol: 206924
Protocol: 206924

Population: Intent-to-Treat

Table 2.2 Summary of Correct Use at Visit 1

| Attempt: 1 | 5-7 Year<br>Stratum<br>(N=xxx) | 8-11 Year<br>Stratum<br>(N=xxx) | Total<br>(N=xxx) |
|---|---|---|---|
| Number of participants who demonstrated correct use Number of participants who did not demonstrate correct use | xxx (xx%)<br>xxx (xx%) | xxx (xx%)<br>xxx (xx%) | xxx (xx%) |
| Reasons for incorrect use [1]: | | | |
| Participant did not slide the cover completely down to expose the mouthpiece until a 'click' is heard | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Participant did shake the inhaler | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Participant did not breathe out (exhales) while holding the inhaler away from their mouth | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Participant did breathe into the mouthpiece | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Participant did not place mouthpiece between lips, and closes firmly around it | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Participant did not take one long steady breath in through their mouth | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Participant did block the air vent with fingers | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Participant did not remove inhaler from his/her mouth and holds his/her breath | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Participant did not breathe out slowly and gently | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Participant did not close the inhaler completely | xxx (xx%) | xxx (xx%) | xxx (xx%) |

Note: Attempts 1, 2 and 3 the Healthcare Professional trains the participant in correct use of the ELLIPTA DPI. Attempts 4 and 5 the parents/guardians assist the participant in demonstrating correct use of the ELLIPTA DPI.

Note: Participants can be counted more than once depending on the reasons for incorrect use.

[1] Percentage for individual incorrect use reasons are calculated based on number of participants who did not demonstrate correct use.

Programming note: Repeat for attempts 2 to 5.


Protocol: 206924 Population: Modified Intent-to-Treat

Table 2.7
Summary of Participants Ease of Use at Visit 2

Questionnaire: Overall

| | | 5-7 Year<br>Stratum<br>(N=xxx) | 8-11 Year<br>Stratum<br>(N=xxx) | Total<br>(N=xxx) |
|---|---|---|---|---|
| Is it easy or hard to use the ELLIPTA inhaler? | n<br>Easy<br>Hard | xxx<br>xxx (xx%)<br>xxx (xx%) | xxx (xx%) | xxx (xx%)<br>xxx (xx%) |
| Is it easy or hard to tell how many puffs are left in the ELLIPTA inhaler? | n | XXX | xxx | xxx |
| | Easy<br>Hard | xxx (xx%)<br>xxx (xx%) | xxx (xx%) | xxx (xx%) |

Programming note: Repeat for "Questionnaire: Version A, Version B"


Example: EFF\_T4
Protocol: 206924

Population: Modified Intent-to-Treat

## Table 2.x Summary of Parent/Guardians Ease of Use at Visit 2

Questionnaire: Overall

| | | Stra | Year<br>atum<br>xx) | St | .1 Year<br>ratum<br>xxx) | Tota<br>(N=x: | |
|---|---|---|---|---|---|---|---|
| Number of parents who attended the final visit also present during the initial training in Correct Use? | n | xxx | | xxx | | xxx | |
| How easy or difficult was it for you to tell how many doses were left in the | n | XXX | | XXX | | XXX | |
| ELLIPTA inhaler? | Verv easv | XXX | (xx%) | XXX | (xx%) | XXX | (xx%) |
| | Easy | XXX | (xx%) | XXX | (xx%) | XXX | (xx%) |
| | Difficult | XXX | (xx%) | XXX | (xx%) | XXX | (xx%) |
| | Very difficult | XXX | (xx%) | XXX | (xx%) | XXX | (xx%) |
| | Very easy/Easy | XXX | (xx%) | XXX | (xx%) | XXX | (xx%) |
| If your child's current inhaled asthma medication was available in the ELLIPTA inhaler, how likely would you be to request | n | xxx | | XXX | | | |
| the ELLIPTA inhaler from your child's doctor? | Very Likely | XXX | (xx%) | XXX | (xx%) | XXX | (xx%) |
| _ | Likely | | (xx%) | | (xx%) | | (xx%) |
| | Unlikely | XXX | (xx%) | XXX | (xx%) | XXX | (xx%) |
| | Very unlikely | XXX | (xx%) | XXX | (xx%) | XXX | (xx%) |
| Programming note: Percet for Wougetienneire. | Very likely/Likely | XXX | (xx%) | XXX | (xx%) | XXX | (xx%) |

Programming note: Repeat for "Questionnaire: Version A, Version B"

Example: EFF\_T5 Protocol: 206924

Population: Modified Intent-to-Treat

Table 2.xx Summary of Protocol Defined Endpoints for Correct Use and Ease of Use at Visit 2 by Age Stratum

| | 5-7 Year | Stratum<br>(N=xxx) | - | | Stratum<br>(N=xxx) |
|---|---|---|---|---|---|
| Number of participants who demonstrate correct use at Visit 2 without assistance from their parents/guardians (Attempt #1) | xx (xx%) | (xx%, xx%) | xx | (xx%) | (xx%, xx%) |
| Number of participants who rate the use of ELLIPTA as easy, among those who demonstrate correct use of the inhaler at Visit 2 [1] | xx (xx%) | (xx%, xx%) | XX | (xx%) | (xx%, xx%) |
| Number of participants who rate the ability to tell how many doses are remaining in the ELLIPTA as easy at Visit 2 | xx (xx%) | (xx%, xx%) | XX | (xx%) | (xx%, xx%) |
| Number of participant's parents/guardians who rate the ability to tell how many doses are remaining in the ELLIPTA as easy or very easy at Visit 2 | xx (xx%) | (xx%, xx%) | XX | (xx%) | (xx%, xx%) |
| Number of participant's parents/guardians who would be likely or very likely to ask their doctor for the ELLIPTA inhaler if the participants current daily inhaled medication(s) were available in the ELLIPTA inhaler | xx (xx%) | (xx%, xx%) | XX | (xx%) | (xx%, xx%) |
| Number of participants who demonstrate correct use at Visit 2 with assistance from their parents/guardians (Attempt #2) | xx (xx%) | (xx%, xx%) | XX | (xx%) | (xx%, xx%) |
| Number of participants who demonstrate correct use at Visit 2 with or without assistance from their parents/guardians (Attempt #1 or Attempt #2) | xx (xx%) | (xx%, xx%) | XX | (xx%) | (xx%, xx%) |

206924

Number of participants who made at least one critical error xx (xx%) (xx%, xx%) xx (xx%) (xx%, xx%) during the use of the ELLIPTA at Visit 2

[1] The percentage is calculated as "number of participants who rate the ELLIPTA as easy" divided by "number of participants who demonstrate correct use at Visit 2 (Attempt #1)" x 100 Note: The 95% CI for the percentages are calculated using the exact binomial distribution.

Programming Note: Please include the following footnotes if any of the composite intercurrent events detailed in the body of the RAP occurred during the study:

For correct use endpoints:

- [#] Denominator used to calculate percentage and precision intervals includes participants who did not fully complete the correct use demonstration and have been deemed as not demonstrating correct use. For questionnaire endpoints:
- [#] Denominator used to calculate percentage and precision include participants who did not answer the question and have been deemed as [not rating the ease of use as easy/not rating the ability to tell how many doses are remaining in the ELLIPTA as easy/not rating the ability to tell how many doses are remaining in the ELLIPTA as Very easy/easy/ not very likely/likely requesting the participant's current daily inhaled medication in the ELLIPTA inhaler]. [Select the ones that apply and write a new footnote for each one]. For critical error endpoint:
- [#] Denominator used to calculate percentage and precision includes participants who did not fully complete all the critical error items in the correct use demonstration and have been deemed as performing a critical error.

206924


Example: EFF\_T6 Protocol: 206924

Population: Modified Intent-to-Treat

### Table 2.15 Summary of Protocol Defined Endpoints for Correct Use and Ease of Use at Visit 2

| | Total<br>(N=xxx) |
|---|---|
| Number of participants who demonstrate correct use at Visit 2 without assistance from their parents/guardians (Attempt #1) | xx (xx%) (xx%, xx%) |
| Number of participants who rate the use of ELLIPTA as easy, among those who demonstrate correct use of the inhaler at Visit 2 [1] | xx (xx%) (xx%, xx%) |
| Number of participants who rate the ability to tell how many doses are remaining in the ELLIPTA as easy at Visit 2 | xx (xx%) (xx%, xx%) |
| Number of participant's parents/guardians who rate the ability to tell how many doses are remaining in the ELLIPTA as easy or very easy at Visit 2 | xx (xx%) (xx%, xx%) |
| Number of participant's parents/guardians who would be likely or very likely to ask their doctor for the ELLIPTA inhaler if the participants current daily inhaled medication(s) were available in the ELLIPTA inhaler | xx (xx%) (xx%, xx%) |
| Number of participants who demonstrate correct use at Visit 2 with assistance from their parents/guardians (Attempt #2) | xx (xx%) (xx%, xx%) |
| Number of participants who demonstrate correct use at Visit 2 with or without assistance from their parents/guardians (Attempt #1 or Attempt #2) | xx (xx%) (xx%, xx%) |

206924

Number of participants who made at least one critical error during the use of the ELLIPTA at Visit  $2\,$ 

xx (xx%) (xx%, xx%)

[1] The percentage is calculated as "number of participants who rate the ELLIPTA as easy" divided by "number of participants who demonstrate correct use at Visit 2 (Attempt #1)" x 100 Note: The 95% CI for the percentages are calculated using the exact binomial distribution.

Programming Note: Please include the following footnotes if any of the composite intercurrent events detailed in the body of the RAP occurred during the study:

For correct use endpoints:

- [#] Denominator used to calculate percentage and precision intervals includes participants who did not fully complete the correct use demonstration and have been deemed as not demonstrating correct use. For questionnaire endpoints:
- [#] Denominator used to calculate percentage and precision include participants who did not answer the question and have been deemed as [not rating the ease of use as easy/not rating the ability to tell how many doses are remaining in the ELLIPTA as easy/ not rating the ability to tell how many doses are remaining in the ELLIPTA as Very easy/easy / not very likely/likely requesting the participant's current daily inhaled medication in the ELLIPTA inhaler]. [Select the ones that apply and write a new footnote for each one]. For critical error endpoint:
- [#] Denominator used to calculate percentage and precision includes participants who did not fully complete all the critical error items in the correct use demonstration and have been deemed as performing a critical error.

206924


Protocol: 206924 Population: Intent-to-Treat

## Table 2.xx Summary of Protocol Defined Endpoints for Correct Use at End of Visit 1 by Age Stratum

| | 5-7 Year Stratum<br>(N=xxx) | 8-11 Year Stratum (N=xxx) |
|---|---|---|
| Number of participants who demonstrate correct use of the ELLIPTA DPI after initial training from the HCP at Visit 1 (Attempt #1) | xx (xx%) (xx%, xx%) | xx (xx%) (xx%, xx%) |
| Number of participants who demonstrate correct use of the ELLIPTA DPI at Visit 1 (Attempt #1 - #5) | xx (xx%) (xx%, xx%) | xx (xx%) (xx%, xx%) |
| Number of participants who made at least one critical error during use of the ELLIPTA DPI after initial training from HCP at Visit 1 (Attempt #1) | xx (xx%) (xx%, xx%) | xx (xx%) (xx%, xx%) |
| Number of participants who made at least one critical error during use of the ELLIPTA DPI at Visit 1 (Attempt #1 - #5) | xx (xx%) (xx%, xx%) | xx (xx%) (xx%, xx%) |

Note: Attempts 1, 2 and 3 the Healthcare Professional trains the participant in correct use of the ELLIPTA DPI. Attempts 4 and 5 the parents/guardians assist the participant in demonstrating correct use of the ELLIPTA DPI.

Note: The 95% CI for the percentages are calculated using the exact binomial distribution.

Programming Note: Please include the following footnotes if any of the composite intercurrent events detailed in the body of the RAP occurred during the study:

For correct use endpoints:

[#] Denominator used to calculate percentage and precision intervals includes participants who did not fully complete the correct use demonstration and have been deemed as not demonstrating correct use. For critical error endpoint:

206924

[#] Denominator used to calculate percentage and precision includes participants who did not fully complete all the critical error items in the correct use demonstration and have been deemed as performing a critical error.

206924

Protocol: 206924

Population: Intent-to-Treat

## Table 2.xx Summary of Protocol Defined Endpoints for Correct Use at End of Visit 1

| | | | Tota<br>(N=xx | | _ |
|---|---|---|---|---|---|
| Number of participants who demonstrate correct use of the ELLIPTA DPI after initial training from the HCP at Visit 1 (Attempt #1) | XX | (xx%) | (xx%, | xx%) | |
| Number of participants who demonstrate correct use of the ELLIPTA DPI at Visit 1 (Attempt #1 - #5) | XX | (xx%) | (xx%, | xx%) | |
| Number of participants who made at least one critical error during use of the ELLIPTA DPI after initial training from the HCP at Visit 1 | XX | (xx%) | (xx%, | xx%) | |
| Number of participants who made at least one critical error during use of the ELLIPTA DPI at Visit 1 (Attempt #1 - #5) | XX | (xx%) | (xx%, | xx%) | |

Note: Attempts 1, 2 and 3 the Healthcare Professional trains the participant in correct use of the ELLIPTA DPI. Attempts 4 and 5 the parents/guardians assist the participant in demonstrating correct use of the ELLIPTA DPI.

Note: The 95% CI for the percentages are calculated using the exact binomial distribution.

Programming Note: Please include the following footnotes if any of the composite intercurrent events detailed in the body of the RAP occurred during the study:

For correct use endpoints:

[#] Denominator used to calculate percentage and precision intervals includes participants who did not fully complete the correct use demonstration and have been deemed as not demonstrating correct use. For critical error endpoint:

206924

[#] Denominator used to calculate percentage and precision includes participants who did not fully complete all the critical error items in the correct use demonstration and have been deemed as performing a critical error.

Example: EFF\_T9
Protocol: 206924

Population: Modified Intent-to-Treat

## Table 2.xx Summary of the Number of Completers of the Ease of Use Questionnaire at Visit 2

Questionnaire: Overall

| | 5-7 Year<br>Stratum<br>(N=xxx) | 8-11 Year<br>Stratum<br>(N=xxx) | Total<br>(N=xxx) |
|---|---|---|---|
| Namban of markining the continue of the continue in | | | |
| Number of participants randomised to an Ease of Use Questionnaire | XXX | XXX | XXX |
| Number of participants who answered the Ease of Use question | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Number of participants who did not answer the Ease of Use question | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Number of participants who answered the number of puffs question | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Number of participants who did not answer the number of puffs question | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Number of participants parents/guardians who answered the number of doses question | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Number of participants parents/guardians who did not answer the number of doses question | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Number of participants parents/guardians who answered the current daily inhaled medication question | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Number of participants parents/guardians who did not answer the current daily inhaled medication question | xxx (xx%) | xxx (xx%) | xxx (xx%) |

Programming note: Repeat for Questionnaire: Version A and Version B

206924


Protocol: 206924 Population: Intent-to-Treat

Table 2.x
Summary of Critical Errors at Visit 1

| Attempt: 1 | 5-7 Year<br>Stratum<br>(N=xxx) | 8-11 Year<br>Stratum<br>(N=xxx) | Total<br>(N=xxx) |
|---|---|---|---|
| Number of participants who performed a critical error | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Number of participants who did not perform a critical error | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Critical errors performed [1]: | | | |
| Participant did not slide the cover completely down to expose the mouthpiece until a 'click' is heard | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Participant did shake the inhaler | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Participant did breathe into the mouthpiece | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Participant did not place mouthpiece between lips, and closes firmly around it | xxx (xx%) | xxx (xx%) | xxx (xx%) |

Note: Attempts 1, 2 and 3 the Healthcare Professional trains the participant in correct use of the ELLIPTA DPI. Attempts 4 and 5 the parents/guardians assist the participant in demonstrating correct use of the ELLIPTA DPI.

Note: Participants can be counted more than once depending on the reasons for critical errors performed. [1] Percentage for individual critical errors performed are calculated based on number of participants who performed a critical error.

Programming note: Repeat for attempts 2 to 5.

206924

Protocol: 206924

Population: Intent-to-Treat

Table 2.xx
Summary of Number of Attempts to Demonstrate Correct Use at Visit 1

| | | 5-7 Year<br>Stratum<br>(N=xxx) | 8-11 Year<br>Stratum<br>(N=xxx) | Total<br>(N=xxx) |
|---|---|---|---|---|
| Number of participants who demonstrated correct use | n | xxx | xxx | xxx |
| Number of participants who did not demonstrate correct | n<br>ise | xxx | xxx | XXX |
| Number of attempts to demonstrate correct use: | n 1 2 3 4 5 Did not demonstrate correct use after 5 attempts | xxx (xx%)<br>xxx (xx%)<br>xxx (xx%)<br>xxx (xx%)<br>xxx (xx%) | xxx (xx%)<br>xxx (xx%)<br>xxx (xx%)<br>xxx (xx%)<br>xxx (xx%) | xxx<br>xxx (xx%)<br>xxx (xx%)<br>xxx (xx%)<br>xxx (xx%)<br>xxx (xx%) |

Note: Attempts 1, 2 and 3 the Healthcare Professional trains the participant in correct use of the ELLIPTA DPI. Attempts 4 and 5 the parents/guardians assist the participant in demonstrating correct use of the ELLIPTA DPI.


Example: EFF\_F1
Protocol: 206924
Population: Intent-to-Treat

Table 2.xx Summary of Correct Use at Visit 1



Note: Attempts 1, 2 and 3 the Healthcare Professional trains the participant in correct use of the ELLIPTA DPI. Attempts 4 and 5 the parents/guardians assist the participant in demonstrating correct use of the ELLIPTA DPI.

Programming Note: Present Age Stratum: 5-7 Year Old, 8-11 Year Old on one page, and Total Population on the second page.

Example: EFF\_F2
Protocol: 206924
Protocol: 206924

Population: Intent-to-Treat

Summary of Ease of Use at Visit 2



Number of Puffs: Responder is defined as the participant's parents/guardians who rate the ability to tell how many doses are remaining in the ELLIPTA as easy or very easy.

Request the ELLIPTA: Responder is defined as the participant's parents/guardians who would be likely or very likely to ask their doctor for the ELLIPTA inhaler if the participants current daily inhaled medication(s) were available in the ELLIPTA inhaler.

Programming Note: Present Age Stratum: 5-7 Year Old, 8-11 Year Old on one page, and Total Population on the second page.

206924

Example: SAFE\_T1 Protocol: 206924

Population: Intent-to-Treat

## Table 3.x Summary of On-Treatment Asthma Exacerbations

| | Total<br>(N=xxx) |
|---|---|
| Number of participants with an Asthma exacerbation | xxx |
| Total number of Asthma exacerbations per participant | |
| n | XXX |
| 0 | xxx (xx%) |
| 1 | xxx (xx%) |
| 2 | xxx (xx%) |
| >=3 | xxx (xx%) |
| Total number of Asthma exacerbations | |
| Total number of exacerbations | XXX |
| Total number of exacerbations leading to a withdrawal from study | xxx |
| Treatment [1][2] | |
| Took oral/systemic corticosteroids | xxx (xx%) |
| Took antibiotics | xxx (xx%) |
| Visited emergency room | xxx (xx%) |
| Hospitalised | xxx (xx%) |
| Intubated | xxx (xx%) |
| Outcome [1] | |
| Resolved | xxx (xx%) |
| Fatal | xxx (xx%) |
| Not resolved | xxx (xx%) |
| | , , |

206924

Example: SAFE\_T1 Page 1 of n
Protocol: 206924

Population: Intent-to-Treat

## Table 3.x Summary of On-Treatment Asthma Exacerbations

| | Total (N=xxx) |
|----------------------------------------|---------------|
| Duration of asthma exacerbation (days) | |
| n | XXX |
| mean | XX.X |
| SD | XX.XX |
| median | XX.X |
| Min. | XX |
| Max. | xx |

<sup>[1]</sup> Percentages calculated using the total number of Asthma exacerbations as the denominator.

<sup>[2]</sup> More than one treatment may be selected for a given exacerbation.

206924

Example: POP\_L1 Protocol: 206924 Page 1 of n

Population: Intent-to-Treat

Listing x
Listing of Treatment Compliance

| Site ID/<br>Unique<br>Subject ID. | Age Stratum | Compliance (%) | Date Placebo<br>Dispensed | Date Placebo<br>Returned | Dose counter start/stop | Total doses<br>Taken |
|---|---|---|---|---|---|---|
| xxxxxx/ | 5-7 Year Old | xx.x | DDMMMYYYY | DDMMMYYYY | 30/xx | xx |

XXXXXX

206924

Example: POP\_L2 Page 1 of n

Protocol: 206924 Population: Intent-to-Treat

## Listing x Listing of Asthma History and Asthma Exacerbation History

Number of exacerbations in the last 12 months that:

Required

| Site ID | Unique<br>Subject ID. | Age Stratum | Asthma Duration | oral/systemic corticosteroid and/or antibiotics [1] | Required hospitalisation |
|---|---|---|---|---|---|
| ×××××× | ×××××× | 5-7 Year Old | <pre>&lt; 1 vear</pre> | x | × |

. . . . .

[1] Not involving hospitalisation

206924


Example: POP\_L3 Protocol: 206924

Population: Intent-to-Treat

# Listing x Listing of Correct Use at Visit 1

| Site ID/<br>Unique<br>Subject ID. | Age Stratum | Date of<br>Assessment/<br>Study Day | Attempt | Demonstrate<br>Correct Use? | Reasons for not demonstrating correct use |
|---|---|---|---|---|---|
| Xxxxxx/<br>Xx | 5-7 Year-Old | DDMMYYYY/<br>1 | 1 | Υ | None |
| Xxxxxx/<br>Xx | 5-7 Year-Old | DDMMYYYY/<br>1 | 1 | N | Participant blocked air vent with fingers |
| | | | 2 | Y | None |

. . . . .

POP\_L4

Protocol: 206924 Page 1 of x

Population: All Subjects Enrolled

## Listing xx Listing of Participants by Country and Site IDs



206924

Example: EFF\_L1
Protocol: 206924

Population: Modified Intent-to-Treat

# Listing x Listing of Correct Use at Visit 2

| Site ID/<br>Unique<br>Subject<br>ID. | Age<br>Stratum | Date of<br>Assessment/<br>Study Day | Questionnaire<br>Version | Attempt | Demonstrate<br>Correct<br>Use? | Reasons for not demonstrating correct use |
|---|---|---|---|---|---|---|
| Xxxxxx/<br>Xx | 5-7<br>Year-Old | DDMMYYYY/<br>27 | Version A | 1 | Y | None |
| Xxxxxx/<br>Xx | 5-7<br>Year-Old | DDMMYYYY/<br>29 | Version B | 1 | N | Participant blocked air vent with fingers |
| | | | | 2 | Y | None |

206924


Example: EFF\_L2 Protocol: 206924

Population: Modified Intent-to-Treat

## Listing x Listing of Ease of Use at Visit 2

| Site ID | Unique<br>Subject ID. | Age<br>Stratum | Visit | Date of<br>Assessment | Study Day | Questionnaire<br>Version | Q1 | Q2 |
|---|---|---|---|---|---|---|---|---|
| Xxxxxx | XXX | 5-7<br>Year-Old | Day 28 | DDMMYYYY | 27 | Version A | Easy | Easy |
| Xxxxxx | xxx | 5-7<br>Year-Old | Day 28 | DDMMYYYY | 29 | Version B | Easy | Hard |

Q1: How easy or difficult (difficult or easy) is it to use the ELLIPTA inhaler?

Q2: How easy or difficult (difficult or easy) is it to tell how many puffs are left in the ELLIPTA inhaler?

206924

Example: SAFE\_L1 Protocol: 206924

Population: Intent-to-Treat


# Listing x Listing of Asthma Exacerbations

| Site ID/<br>Unique<br>Subject ID. | Age Stratum | Date of<br>Onset/<br>Study Day | Date of<br>Resolution/<br>Duration(days) | Severity/<br>Outcome | Withdrawn due<br>to<br>Exacerbation | Systemic or Oral<br>Corticosteroid/<br>Antibiotics | Hospitalised/ Emergency Room/ Intubated/ X-ray performed |
|---|---|---|---|---|---|---|---|
| Xxxxxx/<br>xxxx.xxxx | 5-7 Year-Old | DDMMMYYY/<br>xx | DDMMMYY/<br>xx | Moderate/<br>Recovered/<br>Resolved | N | Y/N | N/N/N |

206924

Example: SAFE\_L2
Protocol: 206924

Protocol: 206924 Page 1 of 1

Population: Intent-to-Treat

Listing x Listing of Deaths

| Site Id./<br>Unique Subject<br>Id. | Age<br>(YEARS)/<br>Sex/<br>Race | Primary Cause of Death | Subreason | Specify | Date of<br>Death/<br>Study Day | Time<br>From<br>Last<br>Dose |
|---|---|---|---|---|---|---|
| PPD | 58/<br>M/<br>WHITE | HAEMORRHAGE | | GASTROINTESTINEL<br>BLEEDING | 2015 <b>PPD</b><br>210 | 9d |